| Print Name & Title | Signature | Date of Signature (DD MMM YYYY) |
|---|---|---|
| Project Manager<br>Dr. Silke Krüger | 115/ | 30 July 2017 |
| Scientist<br>Dr. Jürgen Schrader | i.s.h.m | 30. AUG 2017 |
| Biostatistician<br>Dr. Katharina Ingel | V. Cgo | 30 AUG 2017 |



## **Table of Content**

| Table | e of | Content | 2 |
|-------|------------|---------------------------------------------------|-----|
| 1. | In | troduction | 6 |
| 2. | Ol | bjectives | 7 |
| 3. | In | vestigational Device | 7 |
| 4. | De | esign | 8 |
| 5. | G | eneral Statistical Procedures | 9 |
| 5.1 | | Descriptive analyses | . 9 |
| 5.2 | | Inferential analyses | 10 |
| 5.3 | 3. | Significance level | 10 |
| 5.4 | ٠. | Missing Data | 10 |
| 5.5 | · . | Exclusion of data from confirmatory data analysis | 10 |
| 5.6 | <b>.</b> | Subgroups | 10 |
| 5.7 | <b>'</b> . | Interim analyses | 11 |
| 5.8 | 3. | Software | 11 |
| 6. | Sp | pecific Study Dates | 12 |
| 6.1 | | Enrollment date | |
| 6.2 | | Implantation Date | |
| 6.3 | 3. | Termination Date | 12 |
| 7. | | . , | 13 |
| 7.1 | | Full Analysis Set | |
| 7.2 | | Ilivia Analysis Set | |
| 7.3 | 3. | Plexa Analysis Set | |
| 8. | | | 16 |
| 8.1 | | Analysis set | |
| 8.2 | | Variables | |
| 8.3 | 3. | Treatment of Missing and Spurious Data | |
| 8.4 | ٠. | Exclusion of Particular Information | |
| 8.5 | | Descriptive Analyses | |
| 8.6 | <b>)</b> . | Hypotheses & Statistical Tests | |
| 9. | | | 17 |
| 9.1 | | Analysis set | |
| 9.2 | | Variables | |
| 9.3 | | Treatment of Missing and Spurious Data | |
| 9.4 | | Exclusion of Particular Information | |
| 9.5 | | Descriptive Analyses | |
| 9.6 | | Hypotheses & Statistical Tests | |
| 10. | | • | 20 |
| 10. | | Analysis set | |
| 10. | | Variables | |
| 10. | | Treatment of Missing and Spurious Data | |
| 10. | | Exclusion of Particular Information | |
| 10. | 5. | Descriptive Analyses | 33 |



| 10.6. | Hypotheses & Statistical Tests | 33 |
|--------|------------------------------------------------------------|----|
| 11. PH | HD Data: Ilivia | 34 |
| 11.1. | Analysis set | 34 |
| 11.2. | Variables | 34 |
| 11.3. | Treatment of Missing and Spurious Data | 36 |
| 11.4. | Exclusion of Particular Information | 36 |
| 11.5. | Descriptive Analyses | 36 |
| 11.6. | Hypotheses & Statistical Tests | 36 |
| 12. M | ultipole Pacing Data: Ilivia | 37 |
| 12.1. | Analysis set | 37 |
| 12.2. | Variables | 37 |
| 12.3. | Treatment of Missing and Spurious Data | 43 |
| 12.4. | Exclusion of Particular Information | 43 |
| 12.5. | Descriptive Analyses | 43 |
| 12.6. | Hypotheses & Statistical Tests | 43 |
| 13. Th | nree-month Follow-up Data: Ilivia | 44 |
| 13.1. | Analysis set | 44 |
| 13.2. | Variables | 44 |
| 13.3. | Treatment of Missing and Spurious Data | 46 |
| 13.4. | Exclusion of Particular Information | 46 |
| 13.5. | Descriptive Analyses | 46 |
| 13.6. | Hypotheses & Statistical Tests | 46 |
| 14. Si | x-month Follow-up Data: Ilivia | 47 |
| 14.1. | Analysis set | 47 |
| 14.2. | Variables | 47 |
| 14.3. | Treatment of Missing and Spurious Data | 48 |
| 14.4. | Exclusion of Particular Information | 48 |
| 14.5. | Descriptive Analyses | 48 |
| 14.6. | Hypotheses & Statistical Tests | 48 |
| 15. M | RI Data: Ilivia | 49 |
| 15.1. | Analysis set | 49 |
| 15.2. | Treatment of Missing and Spurious Data | 49 |
| 15.3. | Exclusion of Particular Information | 50 |
| 15.4. | Descriptive Analyses | 50 |
| 15.5. | Hypotheses & Statistical Tests | 50 |
| 16. Pr | rimary Endpoint 1 Ilivia: SADE-free Rate | 51 |
| 16.1. | Analysis set | 51 |
| 16.2. | Variables | 51 |
| 16.3. | Treatment of Missing and Spurious Data | 53 |
| 16.4. | Exclusion of Particular Information | 53 |
| 16.5. | Descriptive Analyses | |
| 16.6. | Hypotheses & Statistical Tests | |
| 16.7. | Alternative analysis (as suggested by the study objective) | 53 |
| 17 54 | econdary FP 1 Ilivia: Vent Arrhythmia Conversion Rate | 54 |



| 17.1. | Analysis set | 54 |
|--------|----------------------------------------|----|
| 17.2. | Variables | 54 |
| 17.3. | Treatment of Missing and Spurious Data | 56 |
| 17.4. | Exclusion of Particular Information | 56 |
| 17.5. | Descriptive Analyses | 56 |
| 17.6. | Hypotheses & Statistical Tests | 56 |
| 18. Ba | aseline Data: Plexa | 57 |
| 18.1. | Analysis Set | 57 |
| 18.2. | Variables | 57 |
| 18.3. | Treatment of Missing and Spurious Data | 59 |
| 18.4. | Exclusion of Particular Information | 59 |
| 18.5. | Descriptive Analyses | 59 |
| 18.6. | Hypotheses & Statistical Tests | 59 |
| 19. In | nplantation Data: Plexa | 60 |
| 19.1. | Analysis set | 60 |
| 19.2. | Variables | 60 |
| 19.3. | Treatment of Missing and Spurious Data | 61 |
| 19.4. | Exclusion of Particular Information | 61 |
| 19.5. | Descriptive Analyses | 61 |
| 19.6. | Hypotheses & Statistical Tests | 61 |
| 20. PH | ID Data: Plexa | 62 |
| 20.1. | Analysis set | 62 |
| 20.2. | Variables | 62 |
| 20.3. | Treatment of Missing and Spurious Data | 62 |
| 20.4. | Exclusion of Particular Information | 62 |
| 20.5. | Descriptive Analyses | 62 |
| 20.6. | Hypotheses & Statistical Tests | 62 |
| 21. Th | ree-month FU Data: Plexa | 63 |
| 21.1. | Analysis set | 63 |
| 21.2. | Variables | 63 |
| 21.1. | Treatment of Missing and Spurious Data | 63 |
| 21.2. | Exclusion of Particular Information | 63 |
| 21.3. | Descriptive Analyses | 63 |
| 21.4. | Hypotheses & Statistical Tests | 63 |
| 22. Si | x-month FU Data: Plexa | 64 |
| 22.1. | Analysis set | 64 |
| 22.2. | Variables | 64 |
| 22.3. | Treatment of Missing and Spurious Data | 64 |
| 22.4. | Exclusion of Particular Information | |
| 22.5. | Descriptive Analyses | 64 |
| 22.6. | Hypotheses & Statistical Tests | |
| 23. Pr | imary Endpoint 2: SADE-free Rate Plexa | 65 |
| 23.1. | Analysis set | 65 |
| 23.2 | Variables | 65 |



| 23.3. | Treatment of Missing and Spurious Data | 67 |
|----------|------------------------------------------------------------|----|
| 23.4. | Exclusion of Particular Information | 67 |
| 23.5. | Descriptive Analyses | 67 |
| 23.6. | Hypotheses & Statistical Tests | 67 |
| 23.7. | Alternative analysis (as suggested by the study objective) | 67 |
| 24. Se | econdary EP: Rate appropriate RV sensing Plexa | 68 |
| 24.1. | Analysis set | 68 |
| 24.2. | Variables | 68 |
| 24.3. | Treatment of Missing and Spurious Data | 68 |
| 24.4. | Exclusion of Particular Information | 68 |
| 24.5. | Descriptive Analyses | 68 |
| 24.6. | Hypotheses & Statistical Tests | 68 |
| 25. Se | econdary EP: Rate appropriate RV pacing Plexa | 69 |
| 25.1. | Analysis set | 69 |
| 25.2. | Variables | 69 |
| 25.3. | Treatment of Missing and Spurious Data | 69 |
| 25.4. | Exclusion of Particular Information | 69 |
| 25.5. | Descriptive Analyses | 69 |
| 25.6. | Hypotheses & Statistical Tests | 69 |
| Abbrevia | ations | 70 |



## 1. Introduction

The aim of this document is to provide detailed instructions on all mandatory descriptive and inferential statistical analyses for the Clinical Investigation Report.

The text contains verbatim excerpts from the CIP. Such excerpts are italicized with grey background; e.g.

This study is designed as post market clinical follow-up study to identify and evaluate residual risks associated with the use of the Ilivia ICD family and the Plexa ICD lead that are unveiled...

The main aspects and the design of the clinical investigation are presented in chapters 2 to 4.

General statistical procedures are summarized in chapter 5. Those methods are used in case there is no other instruction within this document.

Definitions of the specific dates, e.g. effective randomization and termination are presented in chapter 0.

Specific analysis sets are defined in chapter 7.

General data for the complete study are handled in chapter 8. Data related to the Ilivia group and for the Plexa group are handled separately in the subsequent chapters.

Thereby the following statistical considerations are specified:

- Definition of the analysis set for the following analyzes, e.g. excluding patients without any measured or imputed data for this endpoint.
- Definition of the endpoint(s) to be analyzed including references to the source data, e.g. CRF sheet and item.
- Treatment of missing and spurious data for evaluation of the above endpoint(s).
- Exclusion of particular information from the evaluation of the above endpoint(s) in addition to the exclusion of patients from the analysis set.
- Descriptive analyses including tables and figures
- Statistical alternative hypothesis/hypotheses (HA) to analyze the above endpoint(s).
- Statistical tests intended to analyze the above hypothesis/hypotheses.



All variables are defined in tables using the following columns:

Data file Name of a data file exported from the CDMS with one data row per

unique identifier (e.g. patient specific "patient\_display\_ID\_full"). Additionally, a new data file ("data\_SAR") is generated by merging all relevant data from the original CDMS data files and generating derived variables (e.g. BMI from weight and height or date of first AE episode)

Descriptive Information whether data has to be presented with descriptive methods

as defined in the following sub-chapter ("Yes") or data needed for

generating of derived variables only ("No")

Variable name Original name of a variable in the CDMS data file or name of a derived

variables (indicated with a suffix "\_SAR");

note that original labels from the CDMS data will be used

for generating the Statistical Analysis Report unless a new label is

defined in this document ("NEW")

Variable level Nominal, ordinal, scale (metric, continuous), or date Nominal values Values might be shortened ("...") if remaining clear;

note that original values from CDMS data will be used for generating the Statistical Analysis Report unless new nominal values are defined in

this document ("NEW");

for numeric data this information is not applicable (n.a.)

| Data file, unique identifier | Descriptive | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |

# 2. Objectives

#### CIP chapter 7.1 Objectives

This study is designed as post market clinical follow-up study to identify and evaluate residual risks associated with the use of the Ilivia ICD family and the Plexa ICD lead that are unveiled or remained even after risk analysis, risk mitigation and successful conformity assessment. Furthermore, the study aims at providing additional data, as required by regulatory authorities.

# 3. Investigational Device

CIP chapter 4.7. Definition of the investigational Devices

4.7.1 Ilivia ICD family

The Ilivia/Intica/Inlexa ICD family includes the following devices:

- Ilivia 7 VR-T, VR-T DX, DR-T and HF-T QP
- Intica 7 VR-T, VR-T DX, DR-T and HF-T QP
- Intica 5 VR-T, VR-T DX, DR-T
- Inlexa 7 VR-T, VR-T DX, DR-T and HF-T QP
- 4.7.7 Plexa ICD lead



## 4. Design

#### CIP chapter 8. Design of the Clinical Investigation

The study is designed as a multicenter, international, non-randomized, open-label and prospective study including two subgroups: group A with the Ilivia ICD family and group B with the Plexa right ventricular ICD lead. Patients can be enrolled into both groups, if they receive both study devices, see below for more details.

# Group A Ilivia ICD family

#### **Enrollment:**

In group A, a total of 105 patients will be enrolled. With an expected drop-out rate of 10% a minimum number of 94 patients will be included in the analysis set. In total, 26 patients should receive a single chamber ICD, 26 patients a dual chamber ICD and 53 patients a triple chamber ICD (CRT-D).

Tab. 4: Required visit windows (1 month is defined as 30 days)

| | Window | Days post-<br>implant |
|---|---|---|
| Pre-hospital<br>discharge or<br>wound check | + 10 days | 0 to 10 |
| 3 months<br>post-implant | ± 30 days | 61 to 121 |
| 6 months<br>post-implant | ± 30 days | 151 to 211 |

# Group B Plexa ICD lead

#### **Enrollment:**

In group B, a total number of 185 patients will be enrolled. With an expected drop-out rate of 10% a mimimum number of 166 patients will be included in the analysis set.



Fig. 4: Follow-up scheme of group A (Ilivia ICD family) and group B (Plexa ICD lead)



Fig. 5: Overlap of both study groups. Patients implanted with an ICD device of the Ilivia family and a Plexa ICD lead can belong to both groups A and B



## 5. General Statistical Procedures

## 5.1. Descriptive analyses

#### CIP chapter 11.1 Statistical design, methods and analytical procedures

For continuous variables descriptive statistics (mean, standard deviation, minimum, 1. quartile, median, 3. quartile and maximum) will be calculated. For nominal variables absolute numbers and relative frequencies based on the non-missing data will be determined. Ordinal data are described by the 1. quartile, median, and 3. quartile as well as the absolute numbers and relative frequencies based on the non-missing data of each category

Ordinal data are described by the absolute numbers and relative frequencies based on the non-missing data of each category and by the 1.quartile, median and 3. quartile, when appropriate.

For illustration, see the following standard tables based on dummy data.

## Nominal - dichotomous

| Variable label | Category | Missing<br>data | Non-<br>missing<br>data | Absolute frequency | Relative<br>frequency<br>[%] |
|---|---|---|---|---|---|
| Sex | Female | 1 | 9 | 5 | 55.6 |
| History of AF | Yes | 2 | 8 | 4 | 50.0 |

#### Nominal - more than two categories

| NYHA dass,<br>all patients | Absolute<br>frequency | Relative<br>frequency<br>[%] |
|---|---|---|
| NYHA I | 5 | 62.5 |
| NYHA II | 1 | 12.5 |
| NYHA III | 1 | 12.5 |
| NYHA IV | 1 | 12.5 |
| Sum | 8 | 100.0 |

NYHA class, all patients; N total =10; N missing = 2

## Scale / metric

| Variable | N non-<br>missing | N<br>missing | Mean | SD | Min | Lower<br>quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|---|---|---|
| Age [years] | 7 | 3 | 51.7 | 15.0 | 25.0 | 40.0 | 57.0 | 60.0 | 70.0 |
| Height [cm] | 8 | 2 | 177.3 | 14.4 | 150.0 | 170.0 | 179.0 | 187.5 | 195.0 |
| Weight [kg] | 7 | 3 | 77.1 | 14.5 | 55.0 | 69.0 | 77.0 | 90.0 | 99.0 |

#### Ordinal

| Variable | N non-<br>missing | N<br>missing | Min | Lower quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|---|
| NYHA class | 8 | 2 | 1.0 | 1.0 | 1.0 | 2.5 | 4.0 |
| Patient self assessment | 8 | 2 | 1.0 | 1.0 | 1.0 | 2.0 | 3.0 |



## 5.2. Inferential analyses

#### CIP chapter 11.1 Statistical design, method and analytical procedures

For both primary hypotheses exact binomial tests are carried out. All endpoints are analysed per-protocol (PP), whereby the analysis sets are defined for each hypothesis separately.

## 5.3. Significance level

#### CIP chapter 11.3 Level of significance and the power of the study

The 2-sided level of significance is alpha = 2.5% for each alternative hypothesis (1-sided 1.25% significance level). Thus, the 2-sided significance level of the global hypothesis of 5% (1-sided 2.5% significance level) is maintained

## 5.4. Missing Data

#### CIP chapter 11.11 Handling of missing, unused and spurious data

Missing or spurious data will not be imputed.

Spurious data, which were not clarified by the query process before CDMS closure, are indicated. If appropriate, descriptive and inferential analyses are performed both with and without such data.

## 5.5. Exclusion of data from confirmatory data analysis

## CIP chapter 11.12 Exclusion of data from the confirmatory data analysis

If the patient has atrial fibrillation during the device based measurements, the P-wave amplitude and the atrial threshold are not included in the analysis. Protocol deviations in regard to the follow-up schedule will not result in an exclusion of data in the analysis but will be subject to query management.

If the patient has atrial fibrillation during the device based measurements, data are classified as "not measurable: no p-wave visible" in the CRFs.

#### 5.6. Subgroups

#### CIP chapter 11.9 Specification of subgroups

Results of the Ilivia ICD family and the Plexa ICD lead are analysed separately. No further subgroup analysis is planned.



## 5.7. Interim analyses

#### CIP chapter 11.6 Provision of an Interim analysis

In the BIO\MASTER.Ilivia Family / Plexa study no interim analysis is planned to accept the primary alternative hypothesis, e.g. like in a group-sequential design. However, in case of a significant discrepancy of the enrollment periods between both groups, the first group may be analyzed prior to the overall final analysis. This kind of preliminary analysis would not bias the analysis of the other group, as the hypotheses of both groups are analyzed independently. The preliminary analysis of one group (after completion of data collection for this group) would not constitute a multiple interim testing and therefore does not necessitate further statistical adjustment.

Additionally, specific data will be provided to the Australian competent authorities based on a database-freeze planned Q4 2016. This kind of preliminary analysis would not bias the further data because no investigator except the Coordination Investigator will be informed about the results. Except for safety reasons, no instruction for the further conductance of the clinical investigations will be made based on the preliminary analysis.

During the course of the study, some data may be entered in the CDMS with the signature of the investigator missing. Such data are excluded from the analysis. The following tables define which record status values are considered confirmed or not confirmed.

| Variable name | Nominal vales | Variable name | Nominal vales |
|---|---|---|---|
| record_status_text | Record complete Record contains errors Open query Answered query | record_status | 1<br>3<br>1149<br>1150 |

Datasets not confirmed by the investigator

| Variable name | Nominal vales | Variable name | Nominal vales |
|---|---|---|---|
| record_status_text | Investigator signed<br>Monitor approved<br>Record Clean<br>Field Monitor approved | record_status | 1047<br>1051<br>1052<br>1082 |

Datasets confirmed by the investigator<sup>1</sup>

#### 5.8. Software

All analyses will be carried out using validated software, e.g. SAS version 9.4 or upgrades.

<sup>&</sup>lt;sup>1</sup> Note that all data can be changed based on query management before CDMS closure.



# 6. Specific Study Dates

#### 6.1. Enrollment date

#### CIP chapter 8.8.5 Point of enrollment and study termination

The point of enrollment is defined as the date of signature of the informed consent form by the patient. Study related procedures, documentation and collection/following of adverse events will start from this day on.

| Data file, unique identifier patient_display_id_full | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| | name | label | level | values |
| enrollment | dmicdtc | Patient: Date of IC signature | date | n.a. |

## 6.2. Implantation Date

| Data file, unique identifier patient_display_id_full | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|
| implantation_general_data | imp_visdate | Date of implantation of Ilivia and Plexa | date | n.a. |

#### 6.3. Termination Date

#### CIP chapter 8.8.5 Point of enrollment and study termination

The point of study termination is defined as date of 6-month follow-up for patients with regular study termination. For a non-regular study termination, the following rules apply:

- · If none of the investigational devices could successfully be implanted, date of study termination should be the date of the last unsuccessful implantation attempt.
- · In case of replacement or repositioning of the Plexa ICD lead in patients of Group B date of study termination should be date of revision.
- · In case of withdrawal of a patient's consent, date of study termination should be the date of withdrawal of consent.
- · In case of patient death, the date of study termination should be the date of the patient's death.
- · If patient is lost to follow-up, date of termination should be the date of last contact of the physician to the patient.
- · If patient is defined as drop-out patient for any other reason, date of study termination should be the date of latest medical information of the patient (e.g. follow-up, IEGM).



#### **Ilivia Termination Date**

| Data file, identifier patient_display_id_full | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|
| study_termination | end_visdate | Date of study termination | date | n.a. |
| study_termination | end_group_term | Was group participation in one of the groups already terminated before the overall termination date? | nominal | No<br>Yes, group A terminated<br>Yes, group B terminated |
| study_termination | end_group_term_date | Date of group specific termination | date | n.a. |
| data_SAR | enddate_Ilivia_SAR² | Date of Ilivia study termination | date | n.a. |

#### Plexa Termination Date

| Data file, identifier patient_display_id_full | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|
| data_SAR | enddate_Plexa_SAR <sup>3</sup> | Date of Plexa study termination | date | n.a. |

# 7. Analysis Sets

## 7.1. Full Analysis Set

| Data file, identifier patient_display_id_full | Variable name | Variable label | Variable<br>level | Nominal values |
|---|---|---|---|---|
| enrollment | DMSUBIC | Patient has provided written informed consent | nominal | Yes /No |
| data_SAR | analysis_set_full_SAR4 | Full analysis set | nominal | Yes / No |

<sup>2</sup> IF end\_group\_term = Yes, group A terminated THEN enddate\_Ilivia\_SAR = end\_group\_term\_date

ELSE enddate\_Ilivia\_SAR = end\_visdate

<sup>3</sup> IF end\_group\_term = Yes, group B terminated THEN enddate\_Plexa\_SAR = end\_group\_term\_date

ELSE enddate\_Plexa\_SAR = end\_visdate

<sup>4</sup> IF DMSUBIC = Yes

THEN analysis\_set\_full\_SAR = Yes ELSE analysis\_set\_full\_SAR = No



## 7.2. Ilivia Analysis Set

The analysis set Ilivia consists of all patients in group A and in group AB, who met all in- and exclusion criteria. Patients who did not come in contact with any Ilivia device are not included in the analysis set.

| Data file, identifier patient_display_id_full | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|
| enrollment | DMSUBIC | Patient has provided written informed consent | nominal | Yes /No |
| enrollment | TIINCL01 TIINCL02<br>TIINCL03 TIINCL04<br>TIINCL05 TIINCL06 | Inclusion criteria [] | nominal | Yes /No |
| enrollment | TIEXCL01 TIEXCL02<br>TIEXCL03 TIEXCL04<br>TIEXCL05 TIEXCL06<br>TIEXCL07 | Exclusion criteria [] | nominal | Yes /No |
| implantation_gene<br>ral_data | imp_group | Patient Group | | Device of the Ilivia family (group A) Plexa right ventricular lead (group B) Both Ilivia and Plexa (group AB) |
| study_termination | end_early_a | Reason for<br>early study<br>termination | nominal | Implantation of Ilivia ICD family was planned but not performed (patient did not come in contact with the investigational device) [] |
| study_termination | end_early_ab | Reason for early study termination | nominal | Implantation of Ilivia ICD family and Plexa lead were planned but not performed (patient did not come in contact with the investigational devices) [] |
| data_SAR | analysis_set_Ilivia_<br>SAR <sup>5</sup> | Analysis set Ilivia | nominal | Yes / No |

A list of all patients with early drop-out with patient ID, patient group and reason for early study termination will be provided.

THEN analysis\_set\_Ilivia\_SAR = Yes ELSE analysis\_set\_Ilivia\_SAR = No



<sup>5</sup> IF DMSUBIC = Yes AND
TIINCL01 = Yes AND TIINCL02 = Yes AND TIINCL03 = Yes AND
TIINCL04 = Yes AND TIINCL05 = Yes AND TIINCL06 = Yes AND
TIEXCL01 = No AND TIEXCL02 = No AND TIEXCL03 = No AND
TIEXCL04 = No AND TIEXCL05 = No AND TIEXCL06 = No AND TIEXCL07 = No AND
(imp\_group = ... (group A) OR imp\_group = ... (group AB)) AND
end\_early\_a ≠ Implantation of Ilivia ICD family was planned but not performed ... AND
end\_early\_ab ≠ Implantation of Ilivia ICD family and Plexa lead were planned but not performed ...

## 7.3. Plexa Analysis Set

Similar to the definition of the Ilivia analysis set (see chapter 7.2), the Plexa analysis set consists of all patients in group B and in group AB, who met all in- and exclusion criteria. Patients who did not come in contact with any Plexa lead are not included in the analysis set.

| | 1 | | | 1 |
|---|---|---|---|---|
| Data file, identifier | Variable | Variable | Variable | Nominal |
| patient_display_id_full | name | label | level | values |
| enrollment | DMSUBIC | Patient has | nominal | Yes /No |
| | | provided written | | |
| | | informed consent | | |
| enrollment | TIINCL01 TIINCL02 | Inclusion criteria [] | nominal | Yes /No |
| | TIINCL03 TIINCL04 | | | |
| | TIINCL05 TIINCL06 | | | |
| enrollment | TIEXCL01 TIEXCL02 | Exclusion criteria | nominal | Yes /No |
| | TIEXCL03 TIEXCL04 | [] | | · |
| | TIEXCL05 TIEXCL06 | | | |
| | TIEXCL07 | | | |
| implantation gene | imp group | Patient Group | | Device of the Ilivia family (group A) |
| ral_data | | , | | Plexa right ventricular lead (group B) |
| | | | | Both Ilivia and Plexa (group AB) |
| study termination | end early b | Reason for | nominal | Implantation of Plexa lead was planned |
| | | early study | | but not performed (patient did not |
| | | termination | | come in contact with the |
| | | termination | | investigational device) |
| | | | | [] |
| study termination | end early ab | Reason for | nominal | Implantation of Ilivia ICD family and |
| /= | , | early study | | Plexa lead were planned but not |
| | | termination | | performed (patient did not come in |
| | | COMMITTED | | contact with the investigational |
| | | | | devices) |
| | | | | [] |
| data_SAR | analysis_set_Plexa_ | Analysis set Plexa | nominal | Yes / No |
| | SAR <sup>6</sup> | | | |



<sup>&</sup>lt;sup>6</sup> IF DMSUBIC = Yes AND

TIINCL01 = Yes AND TIINCL02 = Yes AND TIINCL03 = Yes AND

TIINCL04 = Yes AND TIINCL05 = Yes AND TIINCL06 = Yes AND

TIEXCL01 = No AND TIEXCL02 = No AND TIEXCL03 = No AND

TIEXCL04 = No AND TIEXCL05 = No AND TIEXCL06 = No AND TIEXCL07 = No AND

<sup>(</sup>imp\_group = ... (group B) OR imp\_group = ... (group AB)) AND

 $end\_early\_b \ \ \neq \ Implantation \ of \ Plexa \ lead \ was \ planned \ but \ not \ performed \ ... \ AND$ 

end\_early\_ab ≠ Implantation of Ilivia ICD family and Plexa lead were planned but not performed ...

THEN analysis\_set\_Plexa\_SAR = Yes

ELSE analysis\_set\_Plexa\_SAR = No

## 8. General data

## 8.1. Analysis set

All analyses are performed for the full analysis  $set^7$ .

#### 8.2. Variables

| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_gene<br>ral_data | Yes | imp_group | Patient<br>Group | nominal | Device of the Ilivia family (group A)<br>Plexa right ventricular lead (group B)<br>Both Ilivia and Plexa (group AB) |

#### Baseline / Demographics

| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| baseline | Yes | bas_age | Age | scale | n.a. |
| baseline | Yes | bas_weight | Weight [kg] | scale | n.a. |
| baseline | Yes | bas_height | Height [cm] | scale | n.a. |
| baseline | Yes | bas_bmi | BMI [kg/m2] | scale | n.a. |
| baseline | Yes | bas_sex | Gender | nominal | Male<br>Female |

The total study duration will be calculated as the total sum of all patients' time between informed consent and termination. If a patient's study participation is terminated earlier for one of the study arms A or B, the later termination date will be used for this patient.

This total study duration will be used to calculate the mortality in deaths per 100 patientyears.

#### Additionally:

- Number of all patients, that signed the informed consent
- Number of patients in the full analysis set, in the Ilivia analysis set (A) and in the Plexa analysis set (B), and number of patients in both the Ilivia and the Plexa analysis set (AB)
- Number of regular terminations (altogether and per group)
- Number of patients with early study termination (split by reason for early termination, altogether and per group)

#### 8.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 8.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

### 8.5. Descriptive Analyses

See general definitions in chapter 5.1.



<sup>&</sup>lt;sup>7</sup> analysis\_set\_full\_SAR = Yes

## 8.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.

## 9. Baseline Data: Ilivia

## 9.1. Analysis set

All analyses are performed for the Ilivia analysis set<sup>8</sup>.

#### 9.2. Variables

#### Baseline / Demographics

| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| baseline | Yes | bas_age | Age | scale | n.a. |
| baseline | Yes | bas_weight | Weight [kg] | scale | n.a. |
| baseline | Yes | bas_height | Height [cm] | scale | n.a. |
| baseline | Yes | bas_bmi | BMI [kg/m2] | scale | n.a. |
| baseline | Yes | bas_sex | Gender | scale | Male / Female |

## **Baseline / Indications**

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| baseline | Yes | bas_heart_<br>disease | Underlying heart disease | nominal | Ischemic<br>Non-ischemic |
| baseline | Yes | bas_indication | ICD indication | nominal | Primary prevention<br>Secondary prevention |
| baseline | Yes | bas_pacing_<br>dependent | Pacemaker-<br>dependency | nominal | Yes / No |
| baseline | Yes | bas_hf | heart failure | nominal | Yes / No |
| baseline | Yes | bas_lbbb | Left BBB | nominal | Yes / No |
| baseline | Yes | bas_rbbb | Right BBB | nominal | Yes / No |
| baseline | Yes | bas_nyha | heart failure status | nominal <sup>9</sup> | NYHA I<br>NYHA II<br>NYHA III<br>NYHA IV |
| baseline | Yes | bas_atrial_<br>rhythm | Current<br>Atrial rhythm | nominal | [] sinus rhythm Sinus bradycardia Sinus Tachycardia Atrial Fibrillation Atrial Flutter Other SVT |
| baseline | Yes | bas_avblock | AV block | nominal | None<br>I°<br>II°<br>III° |
| baseline | Yes | bas_af_type | History of atrial fibrillation (according to ESC guidelines) | nominal | Paroxysmal (usually ≤ 48h) Persistent (> 7 days [] Long-standing persistent [] Permanent (accepted) |

<sup>8</sup> analysis\_set\_Ilivia\_SAR = Yes

 $<sup>^{9}</sup>$  No conversion to ordinal data planned e.g. to calculate Median and inter-quartile range



| | | | | | None |
|---|---|---|---|---|---|
| baseline | Yes | bas_qrs | QRS Duration [ms] | scale | n.a. |
| baseline | No | bas_rr_interval | Mean RR-interval | scale | n.a. |
| baseline | No | bas_heart_rate | mean heart rate | scale | n.a. |
| baseline | Yes | bas_heart_rate_S<br>AR <sup>10</sup> | mean heart rate<br>[bpm] | scale | n.a. |
| baseline | Yes | bas_lvef | LVEF [%] | scale | n.a. |

#### Baseline / Diseases

| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| baseline | Yes | bas_comorb_01 | Hypertension [] | nominal | Yes /No |
| baseline | Yes | bas_comorb_02 | History of TIA / Stroke | nominal | Yes /No |
| baseline | Yes | bas_comorb_03 | Peripheral vascular disease | nominal | Yes /No |
| baseline | Yes | bas_comorb_04 | Asthma or other [] | nominal | Yes /No |
| baseline | Yes | bas_comorb_05 | [] (COPD) | nominal | Yes /No |
| baseline | Yes | bas_comorb_06 | Renal dysfunction | nominal | Yes /No |
| baseline | Yes | bas_comorb_07 | Sleep apnoea | nominal | Yes /No |
| baseline | Yes | bas_comorb_08 | Liver disease | nominal | Yes /No |
| baseline | Yes | bas_comorb_09 | Diabetes mellitus | nominal | Yes /No |
| baseline | Yes | bas_comorb_10 | Anemia | nominal | Yes /No |
| baseline | Yes | bas_comorb_11 | Cancer | nominal | Yes /No |

#### Baseline / Medication

Baseline medication is reported only, whereby "Other" medications, and medication names, are not reported.

| Data file including<br>rows for each<br>medication per<br>patient per date | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| cm_embedded_log | No | CMBLFL | Baseline medication | nominal | Yes / No |
| cm_embedded_log | No | CMCLAS | Medication class | | ACE inhibitors Angiotensin receptor blocker Aldosterone blocker Betablocker (excluding sotalol) Calcium channel blocker Digoxin Statins Diuretics Anticoagulation Antiplatelets Antiarrhythmics Other |

 $<sup>^{10}</sup>$  IF bas\_heart\_rate  $\neq$  missing THEN bas\_heart\_rate\_SAR = bas\_heart\_rate ELSE IF bas\_rr\_interval  $\neq$  missing THEN bas\_heart\_rate\_SAR = 60000 / bas\_rr\_interval



| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| data_SAR | Yes | med01_SAR <sup>11</sup> | ACE inhibitors | nominal | Yes /No |
| data_SAR | Yes | med02_SAR <sup>12</sup> | Angiotensin receptor blocker | nominal | Yes /No |
| data_SAR | Yes | med03_SAR <sup>13</sup> | Aldosterone blocker | nominal | Yes /No |
| data_SAR | Yes | med04_SAR <sup>14</sup> | Betablocker (excluding sotalol) | nominal | Yes /No |
| data_SAR | Yes | med05_SAR <sup>15</sup> | Calcium channel blocker | nominal | Yes /No |
| data_SAR | Yes | med06_SAR <sup>16</sup> | Digoxin | nominal | Yes /No |
| data_SAR | Yes | med07_SAR <sup>17</sup> | Statins | nominal | Yes /No |
| data_SAR | Yes | med08_SAR <sup>18</sup> | Diuretics | nominal | Yes /No |
| data_SAR | Yes | med09_SAR <sup>19</sup> | Anticoagulation | nominal | Yes /No |
| data_SAR | Yes | med10_SAR <sup>20</sup> | Antiplatelets | nominal | Yes /No |
| data_SAR | Yes | med11_SAR <sup>21</sup> | Antiarrhythmics | nominal | Yes /No |
| data_SAR | Yes | med01_02_SAR <sup>22</sup> | ACE inhibitors OR Angiotensin nomina receptor blocker | | Yes /No |

## 9.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 9.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

## 9.5. Descriptive Analyses

See general definitions in chapter 5.1.

#### 9.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.

```
<sup>11</sup> IF CMBLFL = Yes AND any CMCLAS = ACE inhibitors
                                                                 THEN med01 SAR = Yes ELSE med01 SAR = No
<sup>12</sup> IF CMBLFL = Yes AND any CMCLAS = Angiotensin receptor ...
                                                                 THEN med02_SAR = Yes ELSE med02_SAR = No
<sup>13</sup> IF CMBLFL = Yes AND any CMCLAS = Aldosterone blocker
                                                                 THEN med03_SAR = Yes ELSE med03_SAR = No
^{14} IF CMBLFL = Yes AND any CMCLAS = Betablocker \dots
                                                                 THEN med04_SAR= Yes ELSE med04_SAR = No
^{15} IF CMBLFL = Yes AND any CMCLAS = Calcium channel blocker
                                                                 THEN med05_SAR = Yes ELSE med05_SAR = No
^{16} IF CMBLFL = Yes AND any CMCLAS = Digoxin
                                                                 THEN med06_SAR= Yes ELSE med06_SAR = No
^{17} IF CMBLFL = Yes AND any CMCLAS = Statins
                                                                 THEN med07_SAR = Yes ELSE med07_SAR = No
<sup>18</sup> IF CMBLFL = Yes AND any CMCLAS = Diuretics
                                                                 THEN med08_SAR = Yes ELSE med08_SAR = No
^{19} IF CMBLFL = Yes AND any CMCLAS = Anticoagulation
                                                                 THEN med09_SAR = Yes ELSE med09_SAR = No
<sup>20</sup> IF CMBLFL = Yes AND any CMCLAS = Antiplatelets
                                                                 THEN med10_SAR = Yes ELSE med10_SAR = No
^{21} IF CMBLFL = Yes AND any CMCLAS = Antiarrhythmics
                                                                 THEN med11_SAR = Yes ELSE med11_SAR = No
<sup>22</sup> IF CMBLFL = Yes AND any CMCLAS = ACE inhibitors OR
                                                                 THEN med01_02_SAR= Yes
                       any CMCLAS = Angiotensin receptor ...
```

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



ELSE med01 02 SAR = No

# 10. Implantation Data: Ilivia

## 10.1. Analysis set

All analyses are performed for the Ilivia analysis set<sup>23</sup>.

## 10.2. Variables

## Implantation / ICD/CRTD

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>general_data | Yes | imp_category | Study<br>implantation | nominal | De novo CRT-D / ICD implantation Upgrade from pacemaker [] Upgrade from ICD [] Exchange of ICD / CRT-D [] |
| implantation_<br>general_data | Yes | imp_site | Implantation site | nominal | left / right |
| implantation_<br>general_data | Yes | imp_dev_<br>type_other | Device type | nominal | Single chamber ICD<br>Dual Chamber ICD<br>CRT-D |
| implantation_<br>general_data | Yes | imp_dev | Device model | nominal | Ilivia 7<br>[] |
| implantation_<br>general_data | Yes | imp_dev_type | Device type | nominal | VR-T<br>[] |
| implantation_<br>general_data | Yes | imp_connector | Connector type for RV lead | nominal | DF-1 / DF4 |

#### **Implantation / Leads**

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>general_data | No | imp_rv_model | RV lead model | Nominal | Plexa S<br>[] |
| data_SAR | Yes | imp_rv_model_ SAR <sup>24</sup> | RV lead model | Nominal | Plexa<br>Other |

THEN imp\_rv\_model\_SAR = Plexa ELSE imp\_rv\_model\_SAR = other



<sup>&</sup>lt;sup>23</sup> analysis\_set\_Ilivia\_SAR = Yes

<sup>24</sup> IF imp\_rv\_model = Plexa S OR Plexa SD OR Plexa DF-1 S OR Plexa DF-1 S DX

#### Implantation Analyzer Data / RA

| Data file,<br>identifier patient_<br>display_id_full | Descri<br>ptive | Variable<br>name | Variable label<br>NEW prefix added to all labels<br>"Implantation analyzer data, RA: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_data | Yes | imp_ana_ra_amp | Sensing amplitude [mV] | scale | n.a. |
| implantation_<br>analyzer_data | Yes | imp_ana_ra_imp | Pacing impedance $[\Omega]$ | scale | n.a. |
| implantation_<br>analyzer_data | Yes | imp_ana_ra_thresh | Pacing threshold [V] at Pulse width 0.4 ms | scale | n.a. |
| implantation_<br>analyzer_data | No | imp_ana_ra_thresh2 | Pacing threshold [V] | scale | n.a. |
| implantation_<br>analyzer_data | No | imp_ana_ra_pulse | at Pulse width [ms] | scale | n.a. |
| data_SAR | Yes | imp_ana_ra_thresh_0<br>5 <sup>25</sup> | Pacing threshold [V] at Pulse width 0.5 ms | scale | n.a. |

A pacing threshold must always consist of amplitude and duration (pulse width). It is not reasonable to report one without the other.

Here, the CIP requires using 0.4 ms, but it can be expected that other pulse durations were used because different analyzer devices which are being used in the investigational centers have different standard settings.

In the SAP version 1.0 it has been defined that it will be tested during blind review whether a meaningful number of measurements were performed with another pulse duration than 0.4 ms.

This test showed that, in fact, in a meaningful number of threshold measurements, 0.5 ms has been used, but only single or no other values. The same was found for other analyzer threshold measurements at the implantation (RV, LV).

Therefore, thresholds of analyzer measurements will be reported for 0.4 and 0.5 ms pulse duration. Measurements at other pulse duration (if any) will be discarded.

 $<sup>^{25}</sup>$  IF imp\_ana\_ra\_pulse =0.5 THEN imp\_ana\_ra\_thresh\_05 = imp\_ana\_ra\_thresh2



## Implantation Analyzer Data / RA / Not-measured

| Data file,<br>identifier<br>patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_<br>data | No | imp_ana_ra_<br>amp_no | - | nomi<br>nal | Not measurable: P-wave visible but [] Not measurable: No P-wave visible Not done |
| data_SAR | Yes | imp_ana_ra_<br>amp_no_SAR <sup>26</sup> | Implantation analyzer data, RA: Sensing amplitude | nomi<br>nal | Not measurable: P-wave visible but []Measured |
| implantation_<br>analyzer_<br>data | No | imp_ana_ra_<br>imp_no | - | nomi<br>nal | Above range Below range Not measurable: no overdrive pacing Not done |
| data_SAR | Yes | imp_ana_ra_<br>imp_no_SAR <sup>27</sup> | Implantation analyzer data, RA: Pacing impedance | nomi<br>nal | Out of range<br>Measured |
| implantation_<br>analyzer_<br>data | No | imp_ana_ra_<br>thresh_no | - | nomi<br>nal | Not measured at 0.4 ms No capture with maximum output [] Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_ana_ra_<br>thresh_no_SAR | Implantation analyzer<br>data, RA:<br>Pacing threshold | nomi<br>nal | No capture with maximum output []<br>Measured |

<sup>26</sup> IF imp\_ana\_ra\_amp\_no = Not measurable: P-wave visible but ...

THEN imp\_ana\_ra\_amp\_no\_SAR = imp\_ana\_ra\_amp\_no

ELSE IF imp\_ana\_ra\_amp  $\neq$  missing THEN imp\_ana\_ra\_amp\_no\_SAR = Measured

<sup>27</sup> IF imp\_ana\_ra\_imp\_no = Above range OR imp\_ana\_ra\_imp\_no = Below range

THEN imp\_ana\_ra\_imp\_no\_SAR = Out of range



#### Implantation Analyzer Data / RV

| Data file, identifier patient_display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable label<br>NEW prefix added to all labels<br>"Implantation analyzer data, RV: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_data | Yes | imp_ana_rv_amp | Sensing amplitude [mV] | scale | n.a. |
| implantation_<br>analyzer_data | Yes | imp_ana_rv_imp | Pacing impedance $[\Omega]$ | scale | n.a. |
| implantation_<br>analyzer_data | Yes | imp_ana_rv_thresh | Pacing threshold [V] at Pulse width 0.4 ms | scale | n.a. |
| implantation_<br>analyzer_data | No | imp_ana_rv_thresh2 | Pacing threshold [V] | scale | n.a. |
| implantation_<br>analyzer_data | No | imp_ana_rv_pulse | at Pulse width [ms] | scale | n.a. |
| data_SAR | Yes | imp_ana_rv_thresh0 5 <sup>29</sup> | Pacing threshold [V] at Pulse width 0.5 ms | scale | n.a. |

Pacing threshold measurements will be reported for 0.4 and 0.5 ms separately. See the justification above.

#### Implantation Analyzer Data / RV / Not-measured

| Data file, identifier patient_ display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_<br>data | No | imp_ana_rv_<br>amp_no | - | nomi<br>nal | No intrinsic rhythm Amplitude visible but too low to measure During intrinsic rhythm no R-wave visible Not done |
| data_SAR | Yes | imp_ana_rv_<br>amp_no_SAR <sup>30</sup> | Implantation<br>analyzer data, RV:<br>Sensing amplitude | nomi<br>nal | Amplitude visible but too low to measure<br>During intrinsic rhythm no R-wave visible<br>Measured |
| implantation_<br>analyzer_<br>data | No | imp_ana_rv_<br>imp_no | - | nomi<br>nal | Above range Below range Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_ana_rv_<br>imp_no_SAR <sup>31</sup> | Implantation<br>analyzer data, RV:<br>Pacing impedance | nomi<br>nal | Out of range<br>Measured |
| implantation_<br>analyzer_<br>data | No | imp_ana_rv_<br>thresh_no | - | nomi<br>nal | Not measured at 0.4 ms No capture with maximum output [] Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_ana_rv_<br>thresh_no_SAR | Implantation<br>analyzer data, RV:<br>Pacing threshold | nomi<br>nal | No capture with maximum output [] Measured |

<sup>&</sup>lt;sup>29</sup> IF imp\_ana\_rv\_pulse =0.5 THEN imp\_ana\_rv\_thresh\_05 = imp\_ana\_rv\_thresh2



<sup>&</sup>lt;sup>30</sup> IF imp\_ana\_rv\_amp\_no = Amplitude visible ...OR

 $<sup>^{31}</sup>$  IF imp\_ana\_rv\_imp\_no = Above range OR Below range THEN imp\_ana\_rv\_imp\_no\_SAR = Out of range ELSE IF imp\_ana\_rv\_imp  $\neq$  missing THEN imp\_ana\_rv\_imp\_no\_SAR = Measured

#### Implantation Analyzer Data / LV / 7 Sensing Vectors

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable label, NEW prefix added to all labels "Implantation analyzer data, [specification to]: " | Variable<br>level | Nomin<br>al<br>values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_data | Yes | imp_ana_lv_amp_01 | Sensing amplitude [mV] | scale | n.a. |

The above analyses are performed for all 7 vector permutations, respectively:

- 01 LV1 tip to LV2 ring
- 02 LV1 tip to ICD
- 03 LV2 ring to LV3 ring
- 04 LV2 ring to ICD
- 05 LV3 ring to LV4 ring
- 06 LV3 ring to ICD
- 07 LV4 ring to ICD

#### Implantation Analyzer Data / LV / 7 Sensing Vectors / Not-measured

| Data file,<br>identifier patient_<br>display_id_full | Descr<br>iptive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_data | No | imp_ana_lv_svect_<br>no | - | nomi<br>nal | No intrinsic rhythm Amplitude visible but too low to measure During intrinsic rhythm no R-wave visible Not done |
| data_SAR | Yes | imp_ana_lv_svect_<br>no_SAR <sup>33</sup> | Implantation<br>analyzer<br>data: Any LV<br>pacing<br>vector | nomi<br>nal | Amplitude visible but too low to measure<br>During intrinsic rhythm no R-wave visible<br>At least one vector measured |

```
<sup>32</sup> IF
                                                   THEN imp_ana_rv_thresh_no_SAR = imp_ana_rv_thresh_no
        imp_ana_rv_thresh_no = No capture ...
ELSE IF imp_ana_rv_thresh \neq missing
                                                  THEN imp_ana_rv_thresh_no_SAR = Measured
<sup>33</sup> IF imp_ana_lv_svect_no = Amplitude visible but too low to measure
THEN
                   imp_ana_lv_svect_SAR = Amplitude visible but too low to measure
         imp_ana_lv_amp_0j_no = During intrinsic rhythm no R-wave visible
ELSE IF
                   imp_ana_lv_svect_no = During intrinsic rhythm no R-wave visible imp_ana_lv_amp_0j ≠ missing
THEN
ELSE IF any j=1-7 imp_ana_lv_amp_0j
THEN
                   imp_ana_lv_svect_SAR
                                              = At least one vector measured
```



#### <u>Implantation Analyzer Data / LV / 12 Pacing Vectors</u>

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable label, NEW prefix added to all labels "Implantation analyzer data, [specification to]: " | Variable<br>level | Nomin<br>al<br>values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_data | Yes | imp_ana_lv_imp_01 | Pacing impedance $[\Omega]$ | scale | n.a. |
| implantation_<br>analyzer_data | No | imp_ana_lv_thresh_01 | Pacing threshold [V] | scale | n.a. |
| implantation_<br>analyzer_data | No | imp_ana_lv_pulse_01 | at Pulse width [ms] | scale | n.a. |
| data_SAR | Yes | imp_ana_lv_thresh_01_0<br>4 <sup>34</sup> | Pacing threshold [V] at 0.4 ms | scale | n.a. |
| data_SAR | Yes | imp_ana_lv_thresh_01_0 5 <sup>35</sup> | Pacing threshold [V] at 0.5 ms | scale | n.a. |
| implantation_<br>analyzer_data | No | imp_ana_lv_pns_amp_01 | at pacing amplitude [V] | scale | n.a. |
| data_SAR | Yes | imp_ana_lv_pns_amp_01<br>_04 <sup>36</sup> | Phrenic nerve stimulation threshold [V] at 0.4 ms | scale | n.a. |
| data_SAR | Yes | imp_ana_lv_pns_amp_01<br>_05 <sup>37</sup> | Phrenic nerve stimulation threshold [V] at 0.5 ms | scale | n.a. |

Pacing threshold measurements will be reported for 0.4 and 0.5 ms separately. See the justification above.

The above analyses are performed for the following 12 vector permutations, respectively:

- 01 LV1 tip to LV2 ring
- 02 LV1 tip to LV4 ring
- 03 LV1 tip to RV coil
- 04 LV1 tip to ICD
- 05 LV2 ring to LV1 tip
- 06 LV2 ring to LV4 ring
- 07 LV2 ring to RV coil
- 08 LV3 ring to LV2 ring
- 09 LV3 ring to LV4 ring
- 10 LV3 ring to RV coil
- 11 LV4 ring to LV2 ring
- 12 LV4 ring to RV coil

<sup>&</sup>lt;sup>36</sup> IF imp\_ana\_lv\_pulse\_01 = 0.4 THEN imp\_ana\_lv\_pns\_amp\_01\_04 = imp\_ana\_lv\_pns\_amp\_01
<sup>37</sup> IF imp\_ana\_lv\_pulse\_01 = 0.5 THEN imp\_ana\_lv\_pns\_amp\_01\_05 = imp\_ana\_lv\_pns\_amp\_01



<sup>&</sup>lt;sup>34</sup> IF imp\_ana\_lv\_pulse\_01 =0.4 THEN imp\_ana\_lv\_thresh\_01\_04 = imp\_ana\_lv\_thresh\_01

<sup>&</sup>lt;sup>35</sup> IF imp\_ana\_lv\_pulse\_01 =0.5 THEN imp\_ana\_lv\_thresh\_01\_05 = imp\_ana\_lv\_thresh\_01

### Implantation Analyzer Data / LV /12 Pacing Vectors / Not-measured

| Data file,<br>identifier patient_<br>display_id_full | Descr<br>iptive | Variable<br>name | Variable label, NEW prefix added to all labels "Implantation analyzer data, [specification to]: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>analyzer_data | No | imp_ana_lv_<br>imp_01_no | - | nominal | Above range<br>Below range<br>Not done |
| data_SAR | Yes | imp_ana_lv_<br>imp_01_no_SAR <sup>38</sup> | Implantation analyzer data,<br>LV1 tip to LV2 ring:<br>Pacing impedance | nominal | Out of range<br>Measured |
| implantation_<br>analyzer_data | Yes | imp_ana_lv_<br>thresh_01_no | no capture with maximum output possible | nominal | True / False |
| implantation_<br>analyzer_data | Yes | imp_ana_lv_<br>pns_01 | Phrenic nerve stimulation detected | nominal | Yes / No |

The above analyzes are performed for all 12 vector permutations, respectively.

 $<sup>^{38}</sup>$  IF imp\_ana\_lv\_imp\_01\_no  $\,=\,$  Above range OR Below range THEN imp\_ana\_lv\_imp\_01\_no\_SAR  $\,=\,$  Out of range ELSE IF imp\_ana\_lv\_imp\_01  $\,\,\neq\,$  missing  $\,\,$  THEN imp\_ana\_lv\_imp\_01\_no\_SAR  $\,=\,$  Measured



\_

#### Implantation Device Data / RA

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable name | Variable label, NEW prefix added to all labels "Implantation device data, RA:" | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>device_data | Yes | imp_ra_amp | Sensing amplitude [mV] | metric | n.a. |
| implantation_<br>device_data | Yes | imp_ra_imp | Pacing impedance $[\Omega]$ | scale | n.a. |
| implantation_<br>device_data | Yes | imp_ra_thresh | Pacing threshold [V] at Pulse width 0.4 ms | scale | n.a. |

The CIP requires using 0.4 ms pulse width for all RA and RV threshold measurements. However, in the SAP version 1.0 it has been defined that it will be tested during blind review whether a meaningful number of measurements were performed with another pulse duration than 0.4 ms. This test showed that very few or no threshold measurements used other values than 0.4 ms at RA and RV measurements.

Therefore, thresholds of device measurements will be reported for 0.4 ms pulse duration only and measurements at other pulse duration will be discarded.

#### Implantation Device Data / RA / Not-measured

| Data file,<br>identifier patient_<br>display_id_full | Descr<br>iptive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>device_data | No | imp_ra_<br>amp_no | - | nomi<br>nal | Not measurable: P-wave visible but [] Not measurable: No P-wave visible Not done |
| data_SAR | Yes | imp_ra_<br>amp_no_SAR <sup>39</sup> | Implantation<br>device data, RA:<br>Sensing<br>amplitude | nomi<br>nal | Not measurable: P-wave visible but<br>Measured |
| implantation_<br>device_data | No | imp_ra_<br>imp_no | - | nomi<br>nal | Out of range >3000 Out of range <200 Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_ra_<br>imp_no_SAR <sup>40</sup> | Implantation<br>device data, RA:<br>Pacing<br>impedance | nomi<br>nal | Out of range<br>Measured |
| implantation_<br>device_data | No | imp_ra_<br>thresh_no | - | nomi<br>nal | Not measured at 0 .4 ms No capture with 7.5V possible Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_ra_<br>thresh_no_SAR | Implantation<br>device data, RA:<br>Pacing threshold | nomi<br>nal | No capture with 7.5V possible Measured |

ELSE IF  $imp\_ra\_imp$   $\neq missing$  THEN  $imp\_ra\_imp\_no\_SAR$  = Measured



 $<sup>^{39}</sup>$  IF imp\_ra\_amp\_no = Not measurable: P-wave visible but ...THEN imp\_ra\_amp\_no\_SAR = imp\_ra\_amp\_no ELSE IF imp\_ra\_amp  $_{\neq}$  missing THEN imp\_ra\_amp\_no\_SAR = Measured

 $<sup>^{40}</sup>$  IF imp\_ra\_imp\_no = Out of range >3000 OR Out of range <200 THEN imp\_ra\_imp\_no\_SAR = Out of range

<sup>&</sup>lt;sup>41</sup> IF imp\_ra\_thresh\_no = No capture ... THEN imp\_ra\_thresh\_no\_SAR= imp\_ra\_thresh\_no ELSE IF imp\_ra\_thresh ≠ missing THEN imp\_ra\_thresh\_no\_SAR= Measured

## Implantation Device Data / RV

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable name | Variable label, NEW prefix added to all labels "Implantation device data, RV: " | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>device_data | Yes | imp_rv_amp | Sensing amplitude [mV] | scale | n.a. |
| implantation_<br>device_data | Yes | imp_rv_imp | Pacing impedance $[\Omega]$ | scale | n.a. |
| implantation_<br>device_data | Yes | imp_rv_thresh | Pacing threshold [V] at Pulse width 0.4 ms | scale | n.a. |
| implantation_<br>device_data | Yes | imp_rv_shock | Painless shock impedance $[\Omega]$ | scale | n.a. |

Maesurements at other pulse widths than 0.4 ms will be discarded (see above).



#### Implantation Device Data / RV / Not-measured

| Data file,<br>identifier patient_<br>display_id_full | Descr<br>iptive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>device_data | No | imp_rv_<br>amp_no | - | nomi<br>nal | No intrinsic rhythm Amplitude visible but too low to measure During intrinsic rhythm no R-wave visible Not done |
| data_SAR | Yes | imp_rv_<br>amp_no_SAR <sup>42</sup> | Implantation device data, RV: Sensing amplitude | nomi<br>nal | Amplitude visible but too low to measure<br>During intrinsic rhythm no R-wave visible<br>Measured |
| implantation_<br>device_data | No | imp_rv_<br>imp_no | - | nomi<br>nal | Out of range >3000 Out of range <200 Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_rv_<br>imp_no_SAR <sup>43</sup> | Implantation<br>device data, RV:<br>Pacing<br>impedance | nomi<br>nal | Out of range Measured |
| implantation_<br>device_data | No | imp_rv_<br>thresh_no | - | nomi<br>nal | Not measured at 0 .4 ms No capture with 7.5V possible Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_rv_<br>thresh_no_SAR | Implantation<br>device data, RV:<br>Pacing threshold | nomi<br>nal | No capture with 7.5V possible Measured |
| implantation_<br>device_data | No | imp_rv_<br>shock_no | - | | Out of range >150<br>Out of range <25<br>Not done |
| data_SAR | Yes | imp_rv_<br>shock_no_SAR <sup>45</sup> | Implantation<br>device data, RV:<br>Painless shock<br>impedance | nomi<br>nal | Out of range<br>Measured |

42 IF imp\_rv\_amp\_no = Amplitude visible ... OR

 $\begin{array}{lll} imp\_rv\_amp\_no & = During \ intrinsic \dots & THEN \ imp\_rv\_amp\_no\_SAR = imp\_rv\_amp\_no \\ ELSE \ IF \ imp\_rv\_amp & \neq \ missing & THEN \ imp\_rv\_amp\_no\_SAR = Measured \\ \end{array}$ 

<sup>43</sup> IF imp\_rv\_imp\_no = Out of range >3000 OR

 $\begin{array}{lll} imp\_rv\_imp\_no & = Out \ of \ range < 200 & THEN \ imp\_rv\_imp\_no\_SAR & = Out \ of \ range \\ ELSE \ IF \ imp\_rv\_imp & \neq \ missing & THEN \ imp\_rv\_imp\_no\_SAR & = Measured \\ \end{array}$ 

 $^{45}$  IF imp\_rv\_shock\_no = Out of range >150 C



#### Implantation Device Data / LV / 7 Sensing Vectors

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable label, NEW prefix added to all labels "Implantation device data, [specification to]" | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>device_data | Yes | imp_lv_amp_01 | Sensing amplitude [mV] | scale | n.a. |

The above analyses are performed for all 7 vector permutations, respectively:

- 01 LV1 tip to LV2 ring
- 02 LV1 tip to ICD
- 03 LV2 ring to LV3 ring
- 04 LV2 ring to ICD
- 05 LV3 ring to LV4 ring
- 06 LV3 ring to ICD
- 07 LV4 ring to ICD

#### Implantation Device Data / LV / 7 Sensing Vectors / Not-measured

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>device_data | No | imp_lv_<br>svect_no | - | nomi<br>nal | No intrinsic rhythm Amplitude visible but too low to measure During intrinsic rhythm no R-wave visible Not done |
| data_SAR | Yes | imp_lv_<br>svect_SAR <sup>46</sup> | Implantation device data, any LV pacing vector: Sensing amplitude | nomi<br>nal | Amplitude visible but too low to measure<br>During intrinsic rhythm no R-wave visible<br>At least one vector measured |

THEN imp\_lv\_svect\_SAR = Amplitude visible but too low to measure

ELSE IF imp\_lv\_amp\_\_no = During intrinsic rhythm no R-wave visible

imp\_lv\_svect\_SAR = During intrinsic rhythm no R-wave visible THEN

ELSE IF any j=1-7 imp\_lv\_amp\_0j ≠ missing

THEN imp\_lv\_svect\_SAR = At least one vector measured



<sup>&</sup>lt;sup>46</sup> IF = Amplitude visible but too low to measure imp\_lv\_amp\_\_no

#### Implantation Device Data / LV / Programmed Pacing Vectors

Final programmed pacing vectors are handled in the multipole\_pacing CRFs.

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable name | Variable label, NEW prefix added to all labels "Implantation device data, first LV pacing vector: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>device_data | Yes | imp_lv_first_imp | Pacing impedance $[\Omega]$ | scale | n.a. |
| implantation_<br>device_data | No | imp_lv_first_thresh | Pacing threshold [V] | scale | n.a. |
| implantation_<br>device_data | No | imp_lv_first_pulse | at Pulse width [ms] | scale | n.a. |
| data_SAR | Yes | imp_lv_first_thresh_04 <sup>47</sup> | Pacing threshold [V] at Pulse width 0.4 ms | scale | n.a. |

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable name | Variable label, NEW prefix added to all labels "Implantation device data, second LV pacing vector: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>device_data | Yes | imp_lv_sec_imp | Pacing impedance $[\Omega]$ | scale | n.a. |
| implantation_<br>device_data | No | imp_lv_sec_thresh | Pacing threshold [V] | scale | n.a. |
| implantation_<br>device_data | No | imp_lv_sec_pulse | at Pulse width [ms] | scale | n.a. |
| data_SAR | Yes | imp_lv_sec_thresh_04 <sup>48</sup> | Pacing threshold [V] at Pulse width 0.4 ms | scale | n.a. |

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable name | Variable label, NEW prefix added to all labels "Implantation device data, second LV pacing vector: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>device_data | No | imp_lv_first_pvect | Programmed first LV pacing vector | nominal | [] |
| implantation_<br>device_data | No | imp_lv_sec_pvect | Programmed second LV pacing vector | nominal | [] |
| data_SAR | Yes | imp_lv_first_sec_pvect_SA R <sup>49</sup> | Programmed first and second LV pacing vector | nominal | # |

<sup>#</sup> There are 132 possible vector combinations. All vector combinations used in the study have to be reported in the SAR, whereby the most frequent vector combination has to be reported in the CIR, only.

The CIP suggests using 0.4 ms pulse width for all LV threshold measurements, but other values were permitted. In the SAP version 1.0 it has been defined that it will be tested during blind review whether a meaningful number of measurements were performed with another pulse duration than 0.4 ms.

This test showed that very few or no LV threshold measurements used other values than 0.4 ms at implantation.

Therefore, thresholds of device measurements will be reported for 0.4 ms pulse duration only and measurements at other pulse duration will be discarded.

<sup>&</sup>lt;sup>49</sup> imp\_lv\_first\_sec\_pvect\_SAR = combination of imp\_lv\_first\_pvect and imp\_lv\_sec\_pvect per patient



<sup>&</sup>lt;sup>47</sup> IF imp\_lv\_first\_pulse = 0.4, THEN imp\_lv\_first\_thresh\_04 = imp\_lv\_first\_thresh

<sup>&</sup>lt;sup>48</sup> IF imp\_lv\_sec\_pulse = 0.4, THEN imp\_lv\_sec\_thresh\_04 = imp\_lv\_sec\_thresh

#### Implantation Device Data / LV / Programmed Pacing Vectors / Not-measured

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>device_data | No | imp_lv_first_<br>imp_no | - | nomi<br>nal | Out of range >3000 Out of range <200 Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_lv_first_<br>imp_no_SAR <sup>50</sup> | Implantation<br>device data, first<br>LV pacing vector:<br>Pacing impedance | nomi<br>nal | Out of range<br>Measured |
| implantation_<br>device_data | No | imp_lv_first_<br>thresh_no | - | nomi<br>nal | No capture with 7.5V possible<br>Not measurable: no overpacing possible<br>Not done |
| data_SAR | Yes | imp_lv_first_<br>thresh_no_SAR <sup>51</sup> | Implantation<br>device data, first<br>LV pacing vector:<br>Pacing threshold | nomi<br>nal | No capture with 7.5V possible Measured |

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>device_data | No | imp_lv_sec_<br>imp_no | - | nomi<br>nal | Out of range >3000 Out of range <200 Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_lv_sec_<br>imp_no_SAR <sup>52</sup> | Implantation device<br>data, second LV<br>pacing vector:<br>Pacing impedance | nomi<br>nal | Out of range Measured |
| implantation_<br>device_data | No | imp_lv_sec_<br>thresh_no | - | nomi<br>nal | No capture with 7.5V possible Not measurable: no overpacing possible Not done |
| data_SAR | Yes | imp_lv_sec_<br>thresh_no_SAR <sup>53</sup> | Implantation device data, second LV pacing vector: Pacing threshold | nomi<br>nal | No capture with 7.5V possible<br>Measured |



<sup>50</sup> IF imp\_lv\_first\_imp\_no = Out of range > 3000 OR imp\_lv\_first\_imp\_no = Out of range < 200 THEN imp\_l</p>

 $<sup>^{52}</sup>$  IF imp\_lv\_sec\_imp\_no = Out of range >3000 OR imp\_lv\_sec\_imp\_no = Out of range <200 THEN imp\_lv\_sec\_imp\_no\_SAR = Out of range ELSE IF imp\_lv\_sec\_imp  $_{\neq}$  missing THEN imp\_lv\_sec\_imp\_no\_SAR = Measured

## Implantation Device Data / LV / Programmed Delay

| Data file,<br>identifier patient_<br>display_id_full | Descriptive | Variable<br>name | Variable label, NEW prefix added to all labels "Implantation device data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| implantation_<br>device_data | No | imp_order_rvlv | Pacing order | nominal | RV first<br>LV first |
| implantation_<br>device_data | Yes, for the above groups "RV first" and "LV first" | imp_lvlv_delay | LV-LV delay [ms] | scale | n.a. |
| implantation_<br>device_data | Yes, for the above groups "RV first" and "LV first" | imp_rvlv_delay | RV-LV delay [ms] | scale | n.a. |

## 10.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 10.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

### 10.5. Descriptive Analyses

See general definitions in chapter 5.1.

## 10.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



## 11. PHD Data: Ilivia

## 11.1. Analysis set

All analyses are performed for the Ilivia analysis set<sup>54</sup>.

#### 11.2. Variables

#### PHD / General data

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable name | Variable label, NEW prefix added to all labels "PHD data:" | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| phd_general_data | No | phd_visdate | Date of follow-up | date | n.a. |
| phd_general_data | Yes | phd_not_done | visit not performed | nominal | True / False |

The following variables are analyzed as defined for the Ilivia analysis set, as described in chapter 10.2 device data.

PHD Device Data / RA

PHD Device Data / RA / Not-measured

PHD Device Data / RV

PHD Device Data / RV / Not-measured

PHD Device Data / LV / 7 Sensing Vectors

PHD Device Data / LV / 7 Sensing Vectors / Not-measured

PHD Device Data / LV / Programmed Pacing Vectors

PHD Device Data / LV / Programmed Pacing Vectors / Not-measured

Note: all variable names have the prefix "phd\_" instead of "imp\_".

For the programmed first and second LV pacing vector here the pacing threshold should have been measured at pulse width 0.4 ms (phd\_lv\_first\_thresh\_04 and phd\_lv\_sec\_thresh\_04, "Pacing threshold [V] at Pulse width 0.4 ms").

As threshold measurements at other pulse durations than 0.4 will be discarded (see 10.2), the variables "Pacing threshold [V]" (phd\_lv\_first\_thresh and phd\_lv\_sec\_thresh) and "at Pulse width [ms]" (phd\_lv\_first\_pulse and phd\_lv\_sec\_pulse) are not needed for analysis.

However, phd\_lv\_first\_thresh\_no and phd\_lv\_first\_thresh\_no have the additional option "Not measured at 0.4 ms".

<sup>&</sup>lt;sup>54</sup> analysis\_set\_Ilivia\_SAR = Yes





## PHD / Device Data / LV / Vector Change

| Data file,<br>identifier<br>patient_display_id_full | Descriptive | Variable<br>name | Variable label, NEW prefix added to all labels "PHD data: " | Varia<br>ble<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| phd_device_data | Yes | phd_lv_change | Has any of the LV<br>vectors been<br>changed since<br>implant | nomi<br>nal | No Yes, first LV vector Yes, second LV vector Yes, both vectors |
| phd_device_data | Yes | phd_lv_change_<br>reason | Primary reason for change | nomi<br>nal | Phrenic nerve stimulation High LV pacing threshold PNS and high threshold better safety margin [] CRT optimization [] Other |
| phd_device_data | Reporting for each patient if the above variable = other | phd_lv_change_<br>reason_co | [NEW] PHD data:<br>Comments related<br>to Primary reason<br>for change | text | |
| phd_device_data | Yes | phd_lv_change_<br>pns | Phrenic nerve<br>stimulation or high<br>pacing threshold<br>could successfully<br>be resolved | nomi<br>nal | Yes / No |
| phd_device_data | Yes | phd_lv_change_<br>pns_outcome | [New] Actions to resolve PNS | nomi<br>nal | LV lead deactivated<br>Surgical repositioning<br>No action taken<br>Other |
| phd_device_data | Reporting for each patient if the above variable = other | phd_lv_change_<br>pns_co | [NEW] PHD data:<br>Comments related<br>to actions to<br>resolve PNS | text | |

## PHD Device Data / LV Programmed Delay

| Data file,<br>identifier patient_<br>display_id_full | Descriptive | Variable<br>name | Variable label, NEW prefix<br>added to all labels "PHD<br>data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| phd_device_data | Yes | phd_lvlv_reprog | LV-LV delay reprogrammed since implant | nominal | Yes / No |
| phd_device_data | Yes | phd_rvlv_reprog | RV-LV delay reprogrammed since implant | nominal | Yes / No |
| phd_device_data | Yes | phd_order_reprog | Pacing order reprogrammed since implant | nominal | Yes / No |
| phd_device_data | No | phd_order_rvlv | Pacing order | nominal | RV first<br>LV first |
| phd_device_data | Yes, for the above<br>groups "RV first"<br>and "LV first" | phd_lvlv_delay | LV-LV delay [ms] | scale | n.a. |
| phd_device_data | Yes, for the above<br>groups "RV first"<br>and "LV first" | phd_rvlv_delay | RV-LV delay [ms] | scale | n.a. |



## PHD Device Data / CRT / Atrial burden

| Data file,<br>identifier patient_<br>display_id_full | Descr<br>iptive | Variable<br>name | Variable label, NEW prefix added to all labels "PHD data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| phd_device_data | Yes | phd_crt | CRT pacing [%] | scale | n.a. |
| phd_device_data | Yes | phd_aburden | Atrial burden [%] | scale | n.a. |

## 11.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 11.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

## 11.5. Descriptive Analyses

See general definitions in chapter 5.1.

## 11.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.


# 12. Multipole Pacing Data: Ilivia

# 12.1. Analysis set

All analyses are performed for the Ilivia analysis set<sup>55</sup>.

# 12.2. Variables

Multipole Pacing / General Information

| Data file,<br>identifier<br>patient_<br>display_id_full | Descriptive | Variable<br>name | Variable label, NEW prefix added to all labels "Multipole pacing data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | No | mpp_visdate | Date of MPP programming | date | n.a. |
| Multipole_<br>pacing | Yes mpp_visit | | Final programming of<br>MPP has been done | nominal | At implant<br>At Pre-hospital discharge<br>Not done<br>Other |
| Multipole_<br>pacing | Reporting for each patient if the above variable = other | mpp_visit_co | [NEW] Multipole pacing<br>data: Comments<br>related to final<br>programming | text | |
| phd_device_d<br>ata | Yes | phd_lv_first_p<br>vect_no | no LV pacing<br>programmed | nominal | True / False |
| phd_device_d<br>ata | Yes | phd_lv_sec_pv<br>ect_no | no second vector programmed, MPP inactive | nominal | True / False |
| fu_3_month_<br>device_data | Yes | fu3_lv_first_p<br>vect_no | no LV pacing<br>programmed | nominal | True / False |
| fu_3_month_<br>device_data | | | no second vector programmed, MPP inactive | nominal | True / False |
| fu_6_month_<br>device_data | Yes | fu6_lv_first_p<br>vect_no | no LV pacing programmed | nominal | True / False |
| fu_6_month_<br>device_data | Yes | fu6_lv_sec_pv<br>ect_no | no second vector programmed, MPP inactive | nominal | True / False |

A list of all patients with True for one of the "no LV pacing / second vector programmed" variables, together with general comments for the respective follow-up, will be presented.

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



<sup>&</sup>lt;sup>55</sup> analysis\_set\_Ilivia\_SAR = Yes

# Multipole Pacing / LV / Programmed Sensing Vector

| Data file,<br>identifier<br>patient_<br>display_id_full | Descriptive | Variable<br>name | Variable label, NEW prefix added to all labels "Multipole pacing data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | Yes | mpp_lv_svect | Permanent programmed sensing vector | nominal | LV1 tip to LV2 ring [] |
| Multipole_<br>pacing | Yes | mpp_lv_svect_<br>reason | Main reason for vector choice | nominal | Highest amplitude [] Best signal quality Most appropriate [] Standard use of vector Other |
| Multipole_<br>pacing | Reporting for each patient if the above variable = other | mpp_lv_svect_<br>reason_co | [NEW] Multipole pacing data: Comments related to reason for vector choice | text | |



# Multipole Pacing / LV / Programmed Pacing Vectors

| Data file,<br>identifier<br>patient_<br>display_id_full | Descriptive | Variable<br>name | Variable label, NEW prefix added to all labels "Multipole pacing data, first LV pacing vector: " | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | Yes | mpp_lv_<br>first_pvect | Programmed first<br>LV pacing vector | nomi<br>nal | LV1 tip to LV2 ring [] |
| Multipole_<br>pacing | Yes | mpp_lv_<br>first_reason | Main reason for<br>vector choice | nomi<br>nal | According to clinical routine Lowest available threshold To prevent phrenic nerve stimulation Best anatomical position Best available threshold [] According to recommended [] Other |
| Multipole_<br>pacing | Reporting<br>for each pt.<br>if the above<br>variable =<br>other | mpp_lv_<br>first_reason_co | [NEW] Multipole<br>pacing data:<br>Comments related<br>to programmed first<br>vector | text | |

| Data file,<br>identifier<br>patient_<br>display_id_full | Descriptive | Variable<br>name | Variable label, NEW prefix added to all labels "Multipole pacing data, second LV pacing vector: " | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | Yes | mpp_lv_<br>sec_pvect | Programmed second LV pacing vector | nomi<br>nal | [] |
| Multipole_<br>pacing | Yes | mpp_lv_<br>sec_reason | Main reason for vector choice | nomi<br>nal | According to clinical routine Lowest available threshold To prevent phrenic nerve stimulation Best anatomical position Best available threshold [] According to recommended [] Other |
| Multipole_<br>pacing | Reporting<br>for each pt.<br>if the above<br>variable =<br>other | mpp_lv_<br>sec_reason_co | [NEW] Multipole pacing data: Comments related to programmed second vector | text | |
| data_SAR | Yes | mpp_lv_first_se<br>c_pvect_SAR <sup>56</sup> | Programmed first<br>and second LV<br>pacing vector | nomi<br>nal | # |

<sup>\*</sup> A large number of combinations of vector pairs for MPP is possible. Only the most frequent combinations will be reported.

Combinations of two vectors for MPP in which only the designation as "first" and "second" are exchanged will be reported as one.

 $<sup>^{56}</sup>$  mpp\_lv\_first\_sec\_pvect\_SAR = combination of mpp\_lv\_first\_pvect and mpp\_lv\_sec\_pvect per patient



-

### Multipole Pacing / LV / 12 Pacing Vectors

| Data file,<br>identifier patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable label, NEW prefix added to all labels "Multipole pacing data, [specification to]: " | Variable<br>level | Nomin<br>al<br>values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | Yes | mpp_lv_imp_01 | Pacing impedance $[\Omega]$ | scale | n.a. |
| Multipole_<br>pacing | No | mpp_lv_thresh_01 | Pacing threshold [V] | scale | n.a. |
| Multipole_<br>pacing | No | mpp_lv_pulse_01 | at Pulse width [ms] | scale | n.a. |
| data_SAR | Yes | mpp_lv_thresh_01_04 <sup>57</sup> | Pacing threshold [V] at 0.4 ms | scale | n.a. |
| data_SAR | Yes | mpp_lv_thresh_01_15 <sup>58</sup> | Pacing threshold [V] at 1.0 or 1.5 ms | scale | n.a. |
| Multipole_<br>pacing | Yes | mpp_lv_pns_amp_01 | Phrenic nerve stimulation at pacing amplitude [V] | scale | n.a. |

A pacing threshold must always consist of amplitude and duration (pulse width). It is not reasonable to report one without the other.

Here, the CIP does not suggest a specific pulse duration.

In the SAP version 1.0 it has been defined that it will be tested during blind review whether a meaningful number of measurements were performed with another pulse duration than 0.4 ms.

This test showed that most threshold measurements were done with 0.4 ms, but a number were done with 1.0 or 1.5 ms. These will be reported additionally to those at 0.4 ms, because long pulse durations indicate that the threshold was high at shorter pulse durations.

Thresholds of 1.0 and 1.5 ms duration will be summarized because the thresholds at these durations are similar.

The above analyses are performed for the following 12 vector permutations, respectively:

- 01 LV1 tip to LV2 ring
- 02 LV1 tip to LV4 ring
- 03 LV1 tip to RV coil
- 04 LV1 tip to ICD
- 05 LV2 ring to LV1 tip
- 06 LV2 ring to LV4 ring
- 07 LV2 ring to RV coil
- 08 LV3 ring to LV2 ring
- 09 LV3 ring to LV4 ring
- 10 LV3 ring to RV coil
- 11 LV4 ring to LV2 ring12 LV4 ring to RV coil

<sup>58</sup> IF mpp\_lv\_pulse\_01 = 1.0 OR 1.5, THEN mpp\_lv\_thresh\_01\_15 = mpp\_lv\_thresh\_01

BIOTRONII
excellence for life

<sup>&</sup>lt;sup>57</sup> IF mpp\_lv\_pulse\_01 = 0.4, THEN mpp\_lv\_thresh\_01\_04 = mpp\_lv\_thresh\_01

# Multipole Pacing / LV / 12 Pacing Vectors / Not-measured

| Data file,<br>identifier patient_<br>display_id_full | Descr<br>iptive | Variable<br>name | Variable label, NEW prefix added to all labels | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | No | mpp_lv_<br>imp_01_no | - | nominal | Out of range > 3000 out of range < 200 Not done |
| data_SAR | Yes | mpp_lv_<br>imp_01_no SAR <sup>59</sup> | Multipole pacing data,<br>LV1 tip to LV2 ring:<br>Pacing impedance | nominal | Out of range<br>Measured |
| Multipole pacing | No | mpp_lv_thresh_01_n<br>o | - | nominal | True / False |
| data_SAR | Yes | mpp_lv_<br>thresh_01_no_SAR <sup>60</sup> | Multipole pacing data, LV1<br>tip to LV2 ring: Pacing<br>threshold | nominal | No capture with 7.5<br>V possible<br>Measured |
| Multipole_<br>pacing | Yes | mpp_lv_<br>pns_01 | Phrenic nerve stimulation detected | nominal | Yes / No |

The above analyzes are performed for all 12 vector permutations, respectively.

# Multipole Pacing / LV / Programmed Delay

| Data file,<br>identifier patient_<br>display_id_full | Descriptive | Variable<br>name | Variable label,<br>NEW prefix added<br>to all "Multipole<br>pacing data: " | Varia<br>ble<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | Yes | mpp_lvlv_delay_<br>reason | NEW: Main reason<br>for choice of delay<br>LV-LV | nomi<br>nal | According to recommended [] Standard setting used Best hemodynamic response [] Other |
| Multipole_<br>pacing | Yes | mpp_rvlv_delay_<br>reason | NEW: Main reason<br>for choice of delay<br>RV-LV | nomi<br>nal | According to recommended [] Standard setting used Best hemodynamic response [] Other |
| Multipole_<br>pacing | Yes | mpp_order_rvlv | Pacing order | nomi<br>nal | RV first<br>LV first |
| Multipole_<br>pacing | Yes, for<br>the above<br>groups "RV<br>first" and<br>"LV first"" | mpp_lvlv_delay | LV-LV delay [ms] | scale | n.a. |
| Multipole_<br>pacing | Yes, for<br>the above<br>groups "RV<br>first" and<br>"LV first" | mpp_rvlv_delay | RV-LV delay [ms] | scale | n.a. |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



 $<sup>^{59}</sup>$  IF mpp\_lv\_imp\_01\_no = ... > 3000 OR mpp\_lv\_imp\_01\_no = ... < 200 THEN mpp\_lv\_imp\_01\_no\_SAR = Out of range ELSE IF mpp\_lv\_imp\_01  $\neq$  missing THEN mpp\_lv\_imp\_01\_no\_SAR = Measured

 $<sup>^{60}</sup>$  IF <code>mpp\_lv\_thresh\_01\_no</code> = True THEN <code>mpp\_lv\_thres\_01\_no\_SAR=No</code> capture ... ELSE IF <code>mpp\_lv\_thresh\_01</code>  $\neq$  <code>missing</code> THEN <code>mpp\_lv\_thres\_01\_no\_SAR=Measured</code>

# Multipole Pacing / LV /Handling Evaluation

| Data file,<br>identifier<br>patient_<br>display_id_full | Des<br>cript<br>ive | Variable<br>name | Variable label, NEW prefix added to all "Multipole pacing data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | Yes | mpp_handling_activation | Activation of MPP | nominal | Very easy<br>Easy |
| Multipole_<br>pacing | Yes | mpp_handling_navigation | Navigation to MPP programming from the parameter page | nominal | Moderate<br>Moderate-<br>difficult |
| Multipole_<br>pacing | Yes | mpp_handling_lvlv | Programming of LV-LV delay | nominal | Difficult |
| Multipole_<br>pacing | Yes | mpp_handling_rvlv | Programming of RV-LV delay | nominal | |
| Multipole_<br>pacing | Yes | mpp_handling_overall | Overall handling of MPP programmer interface | nominal | |
| data_SAR | Yes | mpp_handling_activation_<br>SAR <sup>61</sup> | Activation of MPP | ordinal | 1/2/3/4/5 |
| data_SAR | Yes | mpp_handling_navigation_<br>SAR <sup>62</sup> | Navigation to MPP programming from the parameter page | ordinal | |
| data_SAR | Yes | mpp_handling_lvlv_<br>SAR <sup>63</sup> | Programming of LV-LV delay | ordinal | |
| data_SAR | Yes | mpp_handling_rvlv_<br>SAR <sup>64</sup> | Programming of RV-LV delay | ordinal | |
| data_SAR | Yes | mpp_handling_overall_<br>SAR <sup>65</sup> | Overall handling of MPP programmer interface | ordinal | |

 $^{61}$  IF mpp\_handling\_activation = Very easy.... THEN mpp\_handling\_activation = 1 ELSE IF mpp\_handling\_activation = Easy.... THEN mpp\_handling\_activation = 2 ELSE IF mpp\_handling\_activation = Moderate.... THEN mpp\_handling\_activation = 3 ELSE IF mpp\_handling\_activation = Moderate-difficult... THEN mpp\_handling\_activation = 4

ELSE IF mpp\_handling\_activation = Difficult

62 see above 63 see above

64 see above 65 see above

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



THEN mpp\_handling\_activation = 5

# Multipole Pacing / LV / Handling Information

| Data file,<br>identifier<br>patient_<br>display_id_full | Des<br>cript<br>ive | Variable<br>name | Variable label, NEW prefix<br>added to all "Multipole<br>pacing data: " | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| Multipole_<br>pacing | Yes | mpp_time_program | At which point in time<br>would you program MPP in<br>a regular CRT-D patient<br>(independent from study<br>set-up) | nomi<br>nal | After implantation Prior to 6 -month FU At 6 -month FU After 6 -month FU Not at all Other |
| Multipole_<br>pacing | Yes | mpp_pat_program | In which patients would you programm MPP? (independent from study participation) | nomi<br>nal | Responder to conventional CRT<br>Non-responder to conventional CRT<br>All CRT patients |
| Multipole_<br>pacing | Yes | mpp_info_sufficient | Did you measure several available vectors during implantation via external analyzer to ensure that sufficient vectors are available due to lead positioning? | nomi<br>nal | Yes / No |
| Multipole_<br>pacing | | mpp_info_sufficient | Was the information sufficient to find suitable vectors for programming later ? | nomi<br>nal | Yes / No |
| Multipole_<br>pacing | Yes | mpp_vect_suitable | Were suitable vectors available for final programming ? | nomi<br>nal | Yes / No |

# 12.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

### 12.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 12.5. Descriptive Analyses

See general definitions in chapter 5.1.

# 12.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 13. Three-month Follow-up Data: Ilivia

# 13.1. Analysis set

All analyses are performed for the Ilivia analysis set<sup>66</sup>.

#### 13.2. Variables

# 3mFU General data

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| fu_3_month_<br>general_data | No | fu3_visdate | Date of 3-month follow-<br>up | date | n.a. |
| fu_3_month_<br>general_data | Yes | fu3_not_done | visit not performed | nominal | True / False |
| fu_3_month_<br>general_data | Yes | fu3_interim | Did another follow-up<br>occur since Pre-hospital<br>discharge | nominal | Yes / No |
| fu_3_month_<br>general_data | Yes | fu3_interim_reason | NEW: Reason for another FU | nominal | Home Monitoring alert<br>Medical symptoms<br>Other |

The following variables are analyzed as defined for the Ilivia analysis set, as described in chapter 11.2.

3mFU Device Data / RA

3mFU Device Data / RA / Not-measured

3mFU Device Data / RV

3mFU Device Data / RV / Not-measured

3mFU Device Data / LV / Programmed Pacing Vectors

3mFU Device Data / LV / Programmed Pacing Vectors / Not-measured

3mFU Device Data / LV / Vector Change

3mFU Device Data / LV / Programmed Delay

3mFU Device Data / CRT / Atrial burden

# 3mFU Device Data / LV / Programmed Sensing Vector

| Data file,<br>identifier<br>patient_<br>display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable label, NEW prefix added to all labels "3m FU data: " | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | Yes | fu3_lv_svect | Permanent programmed sensing vector | nominal | [] |
| fu_3_month_<br>device_data | Yes | fu3_lv_amp | Sensing amplitude [mV] | scale | n.a. |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



<sup>&</sup>lt;sup>66</sup> analysis\_set\_Ilivia\_SAR = Yes

# 3mFU Device Data / LV / Programmed Sensing Vector / Not-measured

| Data file, identifier patient_ display_id_full | Des<br>crip<br>tive | Variable<br>name | Variable<br>label | Varia<br>ble<br>level | Nominal values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | No | fu3_lv_<br>amp_no | - | nomi<br>nal | No intrinsic rhythm Amplitude visible but too low to measure During intrinsic rhythm no R-wave visible Not done |
| data_SAR | Yes | fu3_lv_<br>amp_no_SAR <sup>67</sup> | Implantation device data, any LV pacing vector: Sensing amplitude | nomi<br>nal | Amplitude visible but too low to measure<br>During intrinsic rhythm no R-wave visible<br>Measured |

# 3mFU Device Data / RA /System performance

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | No | fu3_perf_ra_sens | Adequate RA sensing | nominal | Yes / No |
| fu_3_month_<br>devoice_data | Yes | fu3_perf_ra_sens_<br>reason | Reason for inadequate RA sensing | nominal | Oversensing<br>Undersensing<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_ra_pac | Adequate RA pacing | nominal | Yes / No |
| fu_3_month_<br>device_data | Yes | fu3_perf_ra_pac_<br>reason | Reason for inadequate RA pacing | nominal | Non-capture<br>No output<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_ra_pac_<br>nocap | NEW: Reason for non-<br>capture RA | | medical [ ]<br>technical |

# 3mFU Device Data / RV/ System performance

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | No | fu3_perf_rv_sens | Adequate RV sensing | nominal | Yes / No |
| fu_3_month_<br>devoice_data | Yes | fu3_perf_rv_sens_<br>reason | Reason for inadequate RV sensing | nominal | Oversensing<br>Undersensing<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_pac | Adequate RV pacing | nominal | Yes / No |
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_pac_<br>reason | Reason for inadequate RV pacing | nominal | Non-capture<br>No output<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_pac_<br>nocap | NEW: Reason for non-<br>capture RV | | medical [ ]<br>technical |

 $\begin{array}{ccc} & fu3\_lv\_amp\_no & = During \ intrinsic \ rhythm... \ THEN \\ \text{ELSE IF} \ fu3\_lv\_amp & \neq \ missing & THEN \end{array}$ 

fu3\_lv\_amp\_no\_SAR = fu3\_lv\_amp\_no fu3\_lv\_amp\_no\_SAR = Measured

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



<sup>67</sup> IF fu3\_lv\_amp\_no = Amplitude visible ... OR

#### 3mFU Device Data / LV /System performance

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | No | fu3_perf_lv_sens | Adequate LV sensing | nominal | Yes / No |
| fu_3_month_<br>devoice_data | Yes | fu3_perf_lv_sens_<br>reason | Reason for inadequate LV sensing | nominal | Oversensing<br>Undersensing<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_lv_pac | Adequate LV pacing | nominal | Yes / No |
| fu_3_month_<br>device_data | Yes | fu3_perf_lv_pac_<br>reason | Reason for inadequate LV pacing | nominal | Non-capture<br>No output<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_lv_pac_<br>nocap | NEW: Reason for non-<br>capture LV | | medical [ ]<br>technical |

# 13.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

# 13.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 13.5. Descriptive Analyses

See general definitions in chapter 5.1.

# 13.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 14. Six-month Follow-up Data: Ilivia

# 14.1. Analysis set

All analyses are performed for the Ilivia analysis set<sup>68</sup>.

# 14.2. Variables

# 6mFU / General data

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "6mFU data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| fu_6_month_<br>general_data | No | fu6_visdate | Date of 6-month follow-<br>up | date | n.a. |
| fu_6_month_<br>general_data | Yes | fu6_not_done | visit not performed | nominal | True / False |
| fu_6_month_<br>general_data | Yes | fu6_interim | Did another follow-up<br>occur since 3-month<br>Follow-up | nominal | Yes / No |
| fu_6_month_<br>general_data | Yes | fu6_interim_reason | NEW: Reason for another FU | nominal | Home Monitoring alert<br>Medical symptoms<br>Other |

# 6mFU / General Data / Heart Failure

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "6mFU data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| fu_6_month_<br>general_data | No | fu6_hf | Heart failure | nominal | Yes / No |
| fu_6_month_<br>general_data | Yes | fu6_nyha | Heart failure status | nominal | NYHA I<br>NYHA II<br>NYHA III<br>NYHA IV |
| fu_6_month_<br>general_data | Yes | fu6_responder | Responder to CRT-D therapy | nominal | Yes / No |



<sup>&</sup>lt;sup>68</sup> analysis\_set\_Ilivia\_SAR = Yes

The following variables are analyzed as defined for the Ilivia analysis set, as described in chapter 13.2.

6mFU Device Data / RA

6mFU Device Data / RA / Not-measured

6mFU Device Data / RV

6mFU Device Data / RV / Not-measured

6mFU Device Data / LV / Programmed Sensing Vector

6mFU Device Data / LV / Programmed Sensing Vector / Not-measured

6mFU Device Data / LV / Programmed Pacing Vectors

6mFU Device Data / LV / Programmed Pacing Vectors / Not-measured

6mFU Device Data / LV / Vector Change

6mFU Device Data / LV / Programmed Delay

6mFU Device Data / CRT / Atrial burden

# 14.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 14.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 14.5. Descriptive Analyses

See general definitions in chapter 5.1.

### 14.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 15. MRI Data: Ilivia

# 15.1. Analysis set

All analyses are performed for the Ilivia analysis set<sup>69</sup>.

# 3mFU General Data / MRI

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| fu_3_month_<br>general_data | Yes | fu3_mri | Routine MRI scan performed since previous follow-up | nominal | Yes / No |
| fu_3_month_<br>general_data | Yes | fu3_mri_autodetect | MRI AutoDetect feature used or attempted to be used | nominal | Yes / No |

#### 6mFU General Data / MRI

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "6mFU data: " | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| fu_6_month_<br>general_data | Yes | fu6_mri | Routine MRI scan performed since previous follow-up | nominal | Yes / No |
| fu_6_month_<br>general_data | Yes | fu6_mri_autodetect | MRI AutoDetect feature used or attempted to be used | nominal | Yes / No |

# MRI AutoDetect

| Data file, list of<br>MRI events,<br>identifier<br>record_ID | Report all<br>events<br>without any<br>statistics | Variable<br>name | Variable label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| mri_autodetect | Yes | patient_<br>display_id_full | Patient Display ID | nominal | |
| mri_autodetect | Yes | mri_visdate | (Planned) date of MRI scan | nominal | Yes / No |
| mri_autodetect | Yes | mri_successful | MRI AutoDetect could be successfully programmed | nominal | Yes / No |
| mri_autodetect | Yes | mri_test_mode | Was the "MRI Test Mode" used to test the effect of programming the patient to MRI mode? | nominal | Yes / No |
| mri_autodetect | Yes | mri_<br>deactivation_hm | Was deactivation of MRI mode checked via Home Monitoring the day after the scan | nominal | Yes / No |
| mri_autodetect | Yes | mri_ae_dd | Were any Adverse Events/ Device deficiencies detected in regard to the MRI procedure or activation of MRI AutoDetect? | nominal | Yes / No |

# 15.2. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



<sup>69</sup> analysis\_set\_Ilivia\_SAR = Yes

# 15.3. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 15.4. Descriptive Analyses

See general definitions in chapter 5.1.

# 15.5. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 16. Primary Endpoint 1 Ilivia: SADE-free Rate

# 16.1. Analysis set

<u>CIP chapter 11.1. Statistical design, methods and analytical procedures</u>
All endpoints are analysed per-protocol (PP), whereby the analysis sets are defined for each hypothesis separately.

#### CIP chapter 8.1 General considerations

Tab. 4: Required visit windows (1 month is defined as 30 days)

| | Window | Days post-<br>implant |
|--------------------------|-----------|-----------------------|
| 3 months<br>post-implant | ± 30 days | 61 to 121 |

All analyses are performed for a subset of the Ilivia analysis set. To avoid an over-estimation of the SADE-free rate, patients with premature study termination less or equal 60 days after implantation are excluded from the analysis set if no primary endpoint occurred.

#### 16.2. Variables

### CIP chapter 8.3.1.1 Group A: Ilivia family related SADE-free rate through 3 months

The parameter of interest "Ilivia<sub>SADE free</sub>" is the device related SADE-d free rate per patient, which will be calculated by Ilivia<sub>SADE free</sub> = [1 - number of patients with one or more ICD related SADEs (SADE-dI<sub>livia</sub>)until 3-month follow-up divided by all patients in the analysis set] \* 100%. SADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, sport, twiddling) or medical AE caused the SADE, it does not contribute to this endpoint. SADEs that occur later than the 3-months follow-up do not contribute to this endpoint.

In patients without 3 month FU, and in patients with a date of the 3-month Follow-Up outside the required visit window from 61 to 121 days post-implant, all SADEs until and including 121 days after implantation can contribute to the endpoint (if they fulfil the requirements for an endpoint).



| Data file,<br>list of AE evaluations,<br>identifier parent_record_ID | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| ae_evaluation_form_1 | No | endpoint_ilivia →<br>endpoint_ilivia1 | relevant for the primary<br>endpoint (Ilivia family related<br>SADE-free rate) | nominal | Yes / No |
| ae_evaluation_form_1 | No | AESTDT | Onset date | date | n.a. |
| ae_evaluation_form_2 | No | endpoint_ilivia →<br>endpoint_ilivia2 | relevant for the primary<br>endpoint (Ilivia family related<br>SADE-free rate) | nominal | Yes / No |
| ae_evaluation_form_2 | No | AESTDT | Onset date | date | n.a. |

There are two evaluation CRFs. An AE is defined as endpoint relevant when both evaluations came to this result. All divergent evaluations have to be reported<sup>70</sup>.

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_general_<br>data | No | imp_visdate | Date of implantation | date | n.a. |
| data_SAR | No | enddate_Ilivia_SAR | Date of Ilivia study termination | date | n.a. |
| data_SAR | No | date_1stIliviaSADE_SAR <sup>71</sup> | Date of 1 <sup>st</sup> primary<br>Ilivia-related SADE | dummy | No |
| data_SAR | No | Ilivia_primEP_analysis_set_SAR <sup>72</sup> | Analysis set Ilivia primary endpoint | nominal | Yes /No |
| data_SAR | Yes | Ilivia_primEP_SAR <sup>73</sup> | Ilivia-related SADE(s) | nominal | Yes /No |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.

ELSE Ilivia\_primEP\_SAR = No



<sup>&</sup>lt;sup>70</sup> Report any endpoint ilivia1 ≠ endpoint ilivia2

<sup>&</sup>lt;sup>71</sup> date\_1stIliviaSADE\_SAR = minimum AESTDT with endpoint\_ilivia1 = Yes AND endpoint\_ilivia2 = Yes per patient\_display\_id\_full

#### 16.3. Treatment of Missing and Spurious Data

To avoid an over-estimation of the SADE-free rate, patients with premature study termination less or equal 60 days after implantation and without any primary endpoint are excluded from the analysis set.

#### 16.4. Exclusion of Particular Information

All SADEs that occurred later than the 3M-FU, or more than 121 days after implantation, if 3M-FU was outside the required visit window, are not considered.

# 16.5. Descriptive Analyses

Absolute and relative frequencies and additionally the two-sided 97.5% CI are presented.

# 16.6. Hypotheses & Statistical Tests

### CIP chapter 8.3.1.1 Group A: Ilivia family related SADE-free rate through 3 months

Null hypothesis:  $H_{0 \text{ Ilivia}}$ : Ilivia<sub>SADE free</sub>  $\leq 90\%$ 

Alternative hypothesis:  $H_{A\_Ilivia}$ : Ilivia<sub>SADE\_free</sub> > 90%

### CIP chapter 11.1. Statistical design, methods and analytical procedures

For both primary hypotheses exact binomial tests are carried out.

CIP chapter 11.2. Sample size

A correction for multiple testing is considered by adjusting the significance level.

CIP chapter 11.3. Level of significance and the power of the study

The 2-sided level of significance is alpha = 2.5% for each alternative hypothesis (1-sided 1.25% significance level)

A one-sided exact binomial test is carried out for the significance level 1.25%. Additionally, a two-sided 97.5% confidence interval for an exact binomial test is calculated.

# 16.7. Alternative analysis (as suggested by the study objective)

In the definition of the hypothesis, it is stated that endpoints are analyzed if they occur before the 3-months FU (see above, 16.2). However, in section 7 the CIP states that safety through 3 months is the primary study objective.

# 7.1.1 Primary Objectives

# 7.1.1.1 Group A: Ilivia family related safety through 3 months

This objective of the clinical investigation is to confirm the clinical safety of the Ilivia ICD family by the analysis of the Ilivia related SADEs within 3 months after implantation.

A way to analyse the data that is more closely oriented at the study objective than the method described above is a Kaplan-Meyer analysis. The Kaplan-Meyer estimated rate at 91 days represents the best estimate of the target variable.

All patients of the Ilivia analysis set will be included until the time of a first event or censoring due to study discontinuation.



# 17. Secondary EP 1 Ilivia: Vent. Arrhythmia Conversion Rate

# 17.1. Analysis set

<u>CIP chapter 8.3.2.1.1 Percentage of patients with successful fast ventricular arrhythmia conversion by ATP one-shot at 6-month follow-up</u>

This endpoint examines the percentage of patients with successful conversion of ventricular arrhythmia detected in the VF zone by ATP one-shot of all patients with such episodes.

All analyses are performed for patients from the Ilivia analysis set with ventricular arrhythmia episodes detected in the VF zone.

#### 17.2. Variables

<u>CIP chapter 8.3.2.1.1 Percentage of patients with successful fast ventricular arrhythmia conversion by ATP one-shot at 6-month follow-up</u>

This endpoint examines the percentage of patients with successful conversion of ventricular arrhythmia detected in the VF zone by ATP one-shot of all patients with such episodes. Events will only be included in the analysis of this endpoint if

- 1) the arrhythmia was detected in the VF detection zone, and
- 2) if it was classified as true ventricular tachyarrhythmia by the investigator, and
- 3) if ATP one-shot was delivered with the recommended programming (8 pulses with 88% R-S1).

The period under observation starts with the implantation and lasts until the 6-month follow-up. The parameter of interest Conversion  $_{R-S1}$   $_{88\%}$  is defined as following: Conversion  $_{R-S1}$   $_{88\%}$  = (Number of patients with at least one successful conversion / Number of patients with events as defined here) \* 100%.

Thereby, a patient is considered to have experienced successful conversion if at least one episode detected in the VF zone in that patient was converted by ATP one-shot therapies at the recommended programming, i.e ATP one-shot was beneficial and shock delivery could be avoided.

It is possible that ATP one-shot is programmed but not delivered, if the device classifies the rhythm instable. This endpoint will only investigate episodes with delivered ATP one-shot therapy.



| Data file, list of episodes, identifier recoerd_ID | Des<br>crip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| tachyarrhythmia_<br>episode | No | patient_<br>display_id_full | Patient Display ID | nominal | n.a. |
| tachyarrhythmia_<br>episode | No | tac_detect_zone | Detection zone | nominal | nsVT / nsT<br>SVT<br>VT1 / VT2<br>VF |
| tachyarrhythmia_<br>episode | No | tac_assessment | Episode assessment | nominal | non-sustained VT / VF<br>sustained VT / VF<br>SVT / oversensing / other |
| tachyarrhythmia_<br>episode | No | tac_vf_atp_prog | ATP one-shot programming | nominal | 8 pulses with RS1 88%<br>Other programming |
| tachyarrhythmia_<br>episode | No | tac_vf_first_<br>therapy | First therapy attempt | nominal | ATP one-shot<br>Shock |
| tachyarrhythmia_<br>episode | Yes<br># | tac_vf_atp_<br>success | ATP one-shot successfully terminated the episode | nominal | Yes / No |
| dummy | Yes | relevant_secEP_<br>Ilivia_SAR <sup>74</sup> | Episode relevant for secondary endpoint Ilivia | nominal | Yes / No |

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| data_SAR | Yes | Ilivia_secEP_analysis_set_SAR <sup>75</sup> | Analysis set Ilivia secondary endpoint | nominal | Yes /No |
| data_SAR | Yes | Ilivia_secEP_SAR <sup>76</sup> | Any successful ATP<br>(secondary endpoint<br>Ilivia) | nominal | Yes /No |

Beyond the number of patients with endpoint relevant episodes, also the number of episodes, in which ATP-one-shot was delivered (as defined "relevant" in the footnote below) and thereof the number of episodes in which ATP-one-shot was successful (#), will also be reported.

(tac\_assessment = sustained VT / VF OR

tac\_assessment = non-sustained VT / VF ) AND

tac\_vf\_atp\_prog = 8 pulses with RS1 88% AND

tac\_vf\_first\_therapy = ATP one-shot

THEN relevant\_secEP\_Ilivia\_SAR = Yes

ELSE relevant\_secEP\_Ilivia\_SAR = No

<sup>75</sup> IF any relevant\_secEP\_Ilivia\_SAR = Yes per patient\_display\_id\_full

THEN Ilivia\_secEP\_analysis\_set\_SAR = Yes

ELSE Ilivia\_secEP\_analysis\_set\_SAR = No

<sup>76</sup> IF Ilivia\_secEP\_analysis\_set\_SAR = Yes AND

any tac\_vf\_atp\_success = Yes (regarding the relevant episodes) per patient\_display\_id\_full

THEN Ilivia\_secEP\_SAR = Yes

ELSE Ilivia\_secEP\_SAR = No

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



<sup>&</sup>lt;sup>74</sup> IF tac\_detect\_zone = VF AND

# 17.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 17.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 17.5. Descriptive Analyses

See general definitions in chapter 5.1.

# 17.6. Hypotheses & Statistical Tests

<u>CIP chapter 8.3.2.1.1 Percentage of patients with successful fast ventricular arrhythmia conversion by ATP one-shot at 6-month follow-up</u>

No hypotheses are pre-specified for this endpoint due to the low expected number of episodes.

A two-sided 95% confidence interval for an exact binomial test is calculated.



# 18. Baseline Data: Plexa

# 18.1. Analysis Set

All analyses are performed for the Plexa analysis set<sup>77</sup>.

# 18.2. Variables

# Baseline / Demographics

| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| baseline | Yes | bas_age | Age | scale | n.a. |
| baseline | Yes | bas_weight | Weight [kg] | scale | n.a. |
| baseline | Yes | bas_height | Height [cm] | scale | n.a. |
| baseline | Yes | bas_bmi | BMI [kg/m2] | scale | n.a. |
| baseline | Yes | bas_sex | Gender | nominal | Male / Female |

#### Baseline / Indications

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| baseline | Yes | bas_heart_<br>disease | Underlying heart disease | nominal | Ischemic<br>Non-ischemic |
| baseline | Yes | bas_indication | ICD indication | nominal | Primary prevention<br>Secondary prevention |
| baseline | Yes | bas_pacing_<br>dependent | Pacemaker-<br>dependency | nominal | Yes / No |
| baseline | Yes | bas_hf | heart failure | nominal | Yes / No |
| baseline | Yes | bas_lbbb | Left BBB | nominal | Yes / No |
| baseline | Yes | bas_rbbb | Right BBB | nominal | Yes / No |
| baseline | Yes | bas_nyha | heart failure status | nominal <sup>78</sup> | NYHA I ; NYHA II<br>NYHA III ; NYHA IV |
| baseline | Yes | bas_atrial_<br>rhythm | Current<br>Atrial rhythm | nominal | [] sinus rhythm Sinus bradycardia Sinus Tachycardia Atrial Fibrillation Atrial Flutter; Other SVT |
| baseline | Yes | bas_avblock | AV block | nominal | None ; I° ; II° ; III° |
| baseline | Yes | bas_af_type | History of atrial<br>fibrillation<br>(according to ESC<br>guidelines) | nominal | Paroxysmal (usually ≤ 4 8h) Persistent (> 7 days [] Long-standing persistent [] Permanent (accepted) None |
| baseline | Yes | bas_qrs | QRS Duration [ms] | scale | n.a. |
| baseline | No | bas_rr_interval | Mean RR-interval | scale | n.a. |
| baseline | No | bas_heart_rate | mean heart rate | scale | n.a. |
| baseline | Yes | bas_heart_rate_<br>SAR <sup>79</sup> | mean heart rate<br>[bpm] | scale | n.a. |
| baseline | Yes | bas_lvef | LVEF [%] | scale | n.a. |

<sup>77</sup> analysis\_set\_Plexa\_SAR = Yes
78 No conversion to ordinal data planned e.g. to calculate Median and inter-quartile range  $^{79}$  IF bas\_heart\_rate  $\neq$  missing THEN bas\_heart\_rate\_SAR = bas\_heart\_rate ELSE IF bas\_rr\_interval  $\neq$  missing THEN bas\_heart\_rate\_SAR = 60000 / bas\_rr\_interval



# Baseline / Diseases

| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| baseline | Yes | bas_comorb_01 | Hypertension [] | nominal | Yes /No |
| baseline | Yes | bas_comorb_02 | History of TIA / Stroke | nominal | Yes /No |
| baseline | Yes | bas_comorb_03 | Peripheral vascular disease | nominal | Yes /No |
| baseline | Yes | bas_comorb_04 | Asthma or other [] | nominal | Yes /No |
| baseline | Yes | bas_comorb_05 | [] (COPD) | nominal | Yes /No |
| baseline | Yes | bas_comorb_06 | Renal dysfunction | nominal | Yes /No |
| baseline | Yes | bas_comorb_07 | Sleep apnoea | nominal | Yes /No |
| baseline | Yes | bas_comorb_08 | Liver disease | nominal | Yes /No |
| baseline | Yes | bas_comorb_09 | Diabetes mellitus | nominal | Yes /No |
| baseline | Yes | bas_comorb_10 | Anemia | nominal | Yes /No |
| baseline | Yes | bas_comorb_11 | Cancer | nominal | Yes /No |

# **Baseline / Medication**

Baseline medication is reported only, whereby "Other" medications, and medication names, are not reported.

| Data file including<br>rows for each<br>medication per<br>patient per date | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| cm_embedded_log | No | CMBLFL | Baseline medication | nominal | Yes / No |
| cm_embedded_log | No | CMCLAS | Medication class | | ACE inhibitors Angiotensin receptor blocker Aldosterone blocker Betablocker (excluding sotalol) Calcium channel blocker Digoxin Statins Diuretics Anticoagulation Antiplatelets Antiarrhythmics Other |



| Data file, identifier patient_display_id_full | Descrip<br>tive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| data_SAR | Yes | med01_SAR <sup>80</sup> | ACE inhibitors | nominal | Yes /No |
| data_SAR | Yes | med02_SAR <sup>81</sup> | Angiotensin receptor blocker | nominal | Yes /No |
| data_SAR | Yes | med03_SAR <sup>82</sup> | Aldosterone blocker | nominal | Yes /No |
| data_SAR | Yes | med04_SAR <sup>83</sup> | Betablocker (excluding sotalol) | nominal | Yes /No |
| data_SAR | Yes | med05_SAR <sup>84</sup> | Calcium channel blocker | nominal | Yes /No |
| data_SAR | Yes | med06_SAR <sup>85</sup> | Digoxin | nominal | Yes /No |
| data_SAR | Yes | med07_SAR <sup>86</sup> | Statins | nominal | Yes /No |
| data_SAR | Yes | med08_SAR <sup>87</sup> | Diuretics | nominal | Yes /No |
| data_SAR | Yes | med09_SAR <sup>88</sup> | Anticoagulation | nominal | Yes /No |
| data_SAR | Yes | med10_SAR <sup>89</sup> | Antiplatelets | nominal | Yes /No |
| data_SAR | Yes | med11_SAR <sup>90</sup> | Antiarrhythmics | nominal | Yes /No |
| data_SAR | Yes | med01_02_SAR <sup>91</sup> | ACE inhibitors OR Angiotensin receptor blocker | nominal | Yes /No |

# 18.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 18.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 18.5. Descriptive Analyses

See general definitions in chapter 5.1.

### 18.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.

```
<sup>80</sup> IF CMBLFL = Yes AND any CMCLAS = ACE inhibitors
                                                               THEN med01 SAR = Yes ELSE med01 SAR = No
^{\rm 81} IF CMBLFL = Yes AND any CMCLAS = Angiotensin receptor \dots
                                                              THEN med02_SAR = Yes ELSE med02_SAR = No
^{82} IF CMBLFL = Yes AND any CMCLAS = Aldosterone blocker
                                                               THEN med03_SAR = Yes ELSE med03_SAR = No
^{83} IF CMBLFL = Yes AND any CMCLAS = Betablocker ...
                                                               THEN med04_SAR= Yes ELSE med04_SAR = No
^{84} IF CMBLFL = Yes AND any CMCLAS = Calcium channel blocker
                                                               THEN med05_SAR = Yes ELSE med05_SAR = No
85 IF CMBLFL = Yes AND any CMCLAS = Digoxin
                                                               THEN med06_SAR= Yes ELSE med06_SAR = No
^{86} IF CMBLFL = Yes AND any CMCLAS = Statins
                                                               THEN med07_SAR = Yes ELSE med07_SAR = No
<sup>87</sup> IF CMBLFL = Yes AND any CMCLAS = Diuretics
                                                               THEN med08_SAR = Yes ELSE med08_SAR = No
88 IF CMBLFL = Yes AND any CMCLAS = Anticoagulation
                                                              THEN med09_SAR = Yes ELSE med09_SAR = No
89 IF CMBLFL = Yes AND any CMCLAS = Antiplatelets
                                                               THEN med10_SAR = Yes ELSE med10_SAR = No
^{90} IF CMBLFL = Yes AND any CMCLAS = Antiarrhythmics
                                                               THEN med11_SAR = Yes ELSE med11_SAR = No
91 IF CMBLFL = Yes AND any CMCLAS = ACE inhibitors OR
                                                              THEN med01_01_SAR= Yes
                      any CMCLAS = Angiotensin receptor ...
```

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



ELSE med01 02 SAR = No

# 19. Implantation Data: Plexa

# 19.1. Analysis set

All analyses are performed for the Plexa analysis set<sup>92</sup>.

#### 19.2. Variables

#### **General Data**

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_<br>general_data | Yes | imp_rv_model | RV lead model | Nominal | Plexa S<br>Plexa SD<br>Plexa DF-1 S<br>Plexa DF-1 SD<br>Plexa DF-1 S DX<br>[] |
| implantation_<br>general_data | Yes | imp_rv_promri | Pro MRI lead | Nominal | Yes / No |
| implantation_<br>general_data | Yes | imp_rv_length | lead length | Nominal | 60<br>65<br>75<br>60 / 16<br>65 / 16<br>65 / 18<br>75 / 18<br>65 / 15<br>65 / 17 |

The following variables are analyzed as defined for the Ilivia analysis set, as described in chapter 10.2:

Analyzer Data / RA (only Plexa DF-1 S DX)

Analyzer Data / RA / Not-measured (only Plexa DF-1 S DX)

Device Data / RA (only Plexa DF-1 S DX)

Device Data / RA / Not-measured (only Plexa DF-1 S DX)

Analyzer Data / RV

Analyzer Data / RV / Not-measured

Device Data / RV

Device Data / RV / Not-measured

RV measurements will be reported for all Plexa leads, and for Plexa leads with DF4 connectors. Only few leads with DF-1 connector have been implanted, therefore a comparison of the new DF4 connector with historical data may be more reasonable.



<sup>92</sup> analysis\_set\_Plexa\_SAR = Yes

# <u>Handling</u>

| Data file, identifier patient_ display_id_ful | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| plexa_handling | Yes | plx_insertion_site | Insertion site | nominal | L. Subclavian L. Cephalic L. Axillaris R. Subclavian R. Cephalic R. Axillaris |
| plexa_handling | Yes | plx_imp_technique | Implantation technique | nominal | Vein puncture<br>Cutdown |
| plexa_handling | Yes | plx_tip_position | Lead tip position | nominal | RV apex<br>Septal<br>RVOT<br>HIS-bundle<br>Other |
| plexa_handling | Yes | plx_time | Incision to suture time [min] | scale | n.a. |
| plexa_handling | Yes | plx_insertion_assess<br>ment | Lead Insertion Assessment | nominal | Very easy<br>Easy<br>Moderately difficult<br>Difficult |
| plexa_handling | Yes | plx_nb_turns | Number of turns needed to extend the screw | scale | |

# **Handling / Evaluation**

| Data file,<br>identifier patient_<br>display_id_ful | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| plexa_handling | Yes | plx_tracking | Tracking from deployment to target area | nominal | Excellent |
| plexa_handling | Yes | plx_flexibility | Flexibility | nominal | Good<br>Average |
| plexa_handling | Yes | plx_pushability | Pushability | nominal | Fair |
| plexa_handling | Yes | plx_ability_position | Ability to position the lead in the RV | nominal | Poor |
| plexa_handling | Yes | plx_ability_extend | Ability to extend the screw | nominal | |
| plexa_handling | Yes | plx_ability_visualize | Ability to visualize the extended screw | nominal | |
| plexa_handling | Yes | plx_ability_fixate | Ability to fixate the lead tip | nominal | |
| plexa_handling | Yes | plx_radiopacity | Radiopacity in final position | nominal | |

# 19.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 19.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 19.5. Descriptive Analyses

See general definitions in chapter 5.1.

# 19.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



# 20. PHD Data: Plexa

# 20.1. Analysis set

All analyses are performed for the Plexa analysis set<sup>93</sup>.

#### 20.2. Variables

#### PHD / General data

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| phd_general_data | No | phd_visdate | [NEW] Date of PHD | date | n.a. |
| phd_general_data | Yes | phd_not_done | [NEW] PHD:<br>visit not performed | nominal | True / False |

The following variables are analyzed as defined for the Ilivia analysis set, as described in chapter 11.2.

PHD Device Data / RA (only Plexa DF-1 S DX)

PHD Device Data / RA / Not-measured (only Plexa DF-1 S DX)

PHD Device Data / RV

PHD Device Data / RV / Not-measured

RV measurements will be reported for all Plexa leads, and for Plexa leads with DF4 connectors (see 19.2).

# 20.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 20.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

#### 20.5. Descriptive Analyses

See general definitions in chapter 5.1.

# 20.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.

 $<sup>^{93}</sup>$  analysis\_set\_Plexa\_SAR = Yes





# 21. Three-month FU Data: Plexa

# 21.1. Analysis set

All analyses are performed for the Plexa analysis set<sup>94</sup>.

#### 21.2. Variables

The following variables are analyzed as defined for the Ilivia analysis set, as described in chapter 13.2.

3mFU General data

3mFU Device Data / RA (only Plexa DF-1 S DX)

3mFU Device Data / RA / Not-measured (only Plexa DF-1 S DX)

3mFU Device Data / RV

3mFU Device Data / RV / Not-measured

RV measurements will be reported for all Plexa leads, and for Plexa leads with DF4 connectors (see 19.2).

#### 3mFU Device Data / RV/ System performance

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_sens | Adequate RV sensing | nominal | Yes / No |
| fu_3_month_<br>devoice_data | Yes | fu3_perf_rv_sens_<br>reason | Reason for inadequate<br>RV sensing | nominal | Oversensing<br>Undersensing<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_pac | Adequate RV pacing | nominal | Yes / No |
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_pac_<br>reason | Reason for inadequate<br>RV pacing | nominal | Non-capture<br>No output<br>Other |
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_pac_<br>nocap | NEW: Reason for non-<br>capture RV | nominal | medical [ ]<br>technical |

# 21.1. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 21.2. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 21.3. Descriptive Analyses

See general definitions in chapter 5.1.

# 21.4. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses. Note, endpoints with respect to appropriate sensing and pacing at the 3m FU are handled in chapters 24 and 25.

<sup>&</sup>lt;sup>94</sup> analysis set Plexa SAR = Yes





# 22. Six-month FU Data: Plexa

# 22.1. Analysis set

All analyses are performed for the Plexa analysis set<sup>95</sup>.

#### 22.2. Variables

The following variables are analyzed as defined for the Ilivia analysis set, as described in chapter 14.2.

6mFU General data

6mFU Device Data / RA (only Plexa DF-1 S DX)

6mFU Device Data / RA / Not-measured (only Plexa DF-1 S DX)

6mFU Device Data / RV

6mFU Device Data / RV / Not-measured

RV measurements will be reported for all Plexa leads, and for Plexa leads with DF4 connectors (see 19.2).

# 22.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

### 22.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 22.5. Descriptive Analyses

See general definitions in chapter 5.1.

# 22.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.

<sup>95</sup> analysis\_set\_Plexa\_SAR = Yes





# 23. Primary Endpoint 2: SADE-free Rate Plexa

# 23.1. Analysis set

All analyses are performed for the Plexa analysis set <sup>96</sup>.

CIP chapter 11.1 Statistical design, methods and analytical procedures

All endpoints are analysed per-protocol (PP), whereby the analysis sets are defined for each hypothesis separately.

#### CIP chapter 8.1 General considerations

Tab. 4: Required visit windows (1 month is defined as 30 days)

| | Window | Days post-<br>implant |
|-----------------------|-----------|-----------------------|
| 3 months post-implant | ± 30 days | 61 to 121 |

All analyses are performed for a subset of the Plexa analysis set. To avoid an over-estimation of the SADE-free rate, patients with premature study termination less or equal 60 days after implantation are excluded from the analysis set if no primary endpoint occurred.

#### 23.2. Variables

CIP chapter 8.3.1.2 Group B: Plexa related SADE-free rate through 3 months

The parameter of interest "Plexa<sub>SADE free</sub>" is the SADE-free rate per patient, which will be calculated by Plexa <sub>SADE free</sub> = [1 - number of patients with one or more Plexa-related SADEs (SADE-d <sub>Plexa</sub>) until 3-month follow-up divided by all patients in the analysis set] \* 100%. SADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, sport, twiddling) or medical AE caused the SADE, it does not contribute to this endpoint. SADEs that occur later than the 3-months follow-up do not contribute to this endpoint.

In patients without 3M FU and in patients with the 3-months FU outside the CIP defined period, all SADEs until and including 121 days after implantation can contribute to the endpoint (if they fulfil the requirements for an endpoint).



<sup>96</sup> analysis\_set\_Plexa\_SAR = Yes

| Data file,<br>list of AE evaluations,<br>identifier parent_record_ID | Descr<br>iptive | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| ae_evaluation_form_1 | No | endpoint_plexa →<br>endpoint_plexa1 | relevant for the primary<br>endpoint (Plexa related SADE-<br>free rate) | nominal | Yes / No |
| ae_evaluation_form_1 | No | AESTDT | Onset date | date | n.a. |
| ae_evaluation_form_2 | No | endpoint_plexa →<br>endpoint_plexa2 | relevant for the primary<br>endpoint (Plexa related SADE-<br>free rate) | nominal | Yes / No |
| ae_evaluation_form_2 | No | AESTDT | Onset date | date | n.a. |

There are two evaluation CRFs. An AE is defined as endpoint relevant when both evaluations came to this result. All divergent evaluations have to be reported<sup>97</sup>.

| Data file, identifier patient_display_id_full | Descr<br>iptive | Variable name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| implantation_general_<br>data | Yes | imp_visdate | Date of implantation | date | n.a. |
| data_SAR | Yes | enddate_Plexa_SAR | Date of Plexa study termination | date | n.a. |
| data_SAR | No | date_1stPlexaSADE_SAR <sup>98</sup> | Date of 1 <sup>st</sup> primary<br>Plexa-related SADE | dummy | No |
| data_SAR | No | Plexa_primEP_analysis_set_SAR <sup>99</sup> | Analysis set Plexa primary endpoint | nominal | Yes /No |
| data_SAR | Yes | Plexa_primEP_SAR <sup>100</sup> | Plexa-related SADE(s) | nominal | Yes /No |

```
99 IF analysis_set_Plexa_SAR = Yes AND date_1stPlexaSADE_SAR - imp_visdate ≤ 60 days OR enddate_Plexa_SAR - imp_visdate ≥ 61 days
THEN Plexa_primEP_analysis_set_SAR = Yes
ELSE Plexa_primEP_analysis_set_SAR = No

100 IF analysis_set_Plexa_SAR = Yes AND date_1stPlexaSADE_SAR ≠ missing AND {[fu3_visdate ≠ missing AND fu3_visdate is compliant AND date_1stPlexa_SADE_SAR ≤ fu3_visdate] OR [fu3_visdate ≠ missing AND fu3_visdate is not compliant AND date_1stPlexaSADE_SAR - imp_visdate ≤ 121 days] OR [fu3_visdate = missing AND date_1stPlexaSADE_SAR - imp_visdate ≤ 121 days] }
THEN Plexa_primEP_SAR = Yes
```

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.

ELSE Plexa\_primEP\_SAR = No



 $<sup>^{97}</sup>$  Report any endpoint\_plexa1  $\neq$  endpoint\_plexa2

<sup>98</sup> date\_1stPlexaSADE\_SAR = minimum AESTDT with endpoint\_plexa1 = Yes AND endpoint\_plexa2 = Yes per patient\_display\_id\_full

#### 23.3. Treatment of Missing and Spurious Data

To avoid an over-estimation of the SADE-free rate, patients with premature study termination less or equal 60 days after implantation and without any primary endpoint are excluded from the analysis set.

#### 23.4. Exclusion of Particular Information

All SADEs that occurred later than the 3M-FU, or more than 121 days after implantation, if 3M-FU was outside the required visit window, are not considered.

# 23.5. Descriptive Analyses

Absolute and relative frequencies and additionally the two-sided 97.5% CI are presented.

# 23.6. Hypotheses & Statistical Tests

### CIP chapter 8.3.1.1 Group A: Ilivia family related SADE-free rate through 3 months

Null hypothesis:  $H_{0\_Plexa}$ : Plexa<sub>SADE free</sub>  $\leq 90\%$ 

Alternative hypothesis: HA Plexa: PlexaSADE free > 90%

# CIP chapter 11.1. Statistical design, methods and analytical procedures

For both primary hypotheses exact binomial tests are carried out.

CIP chapter 11.2. Sample size

A correction for multiple testing is considered by adjusting the significance level.

CIP chapter 11.3. Level of significance and the power of the study

The 2-sided level of significance is alpha = 2.5% for each alternative hypothesis (1-sided 1.25% significance level)

A one-sided exact binomial test is carried out for the significance level 1.25%. Additionally, a two-sided 97.5% confidence interval for an exact binomial test is calculated.

#### 23.7. Alternative analysis (as suggested by the study objective)

In the definition of the hypothesis, it is stated that endpoints are analyzed if they occurr before the 3-months FU (see above, 23.2). However, in section 7 the CIP states that saftey through 3 months is the primary study objective.

### 7.1.1 Primary Objectives

...

#### 7.1.1.2 Group B: Plexa related safety through 3 months

This objective of the clinical investigation is to confirm the clinical safety of the Plexa ICD lead by the analysis of the Plexa related SADEs within 3 months after implantation.

A way to analyse the data that is more closely oriented at the study objective than the method described above is a Kaplan-Meyer analysis. The Kaplan-Meyer estimated rate at 91 days represents the best estimate of the target variable.

All patients of the Plexa analysis set will be included until the time of a first event or censoring due to study discontinuation.



# 24. Secondary EP: Rate appropriate RV sensing Plexa

# 24.1. Analysis set

All analyses are performed for the Plexa analysis set<sup>101</sup>.

CIP chapter 11.1 Statistical design, methods and analytical procedures

All endpoints are analysed per-protocol (PP), whereby the analysis sets are defined for each hypothesis separately.

#### CIP chapter 8.3.2.2.1 Rate of appropriate right ventricular sensing at 3-month follow-up

Only the evaluation of the 3-month follow-up is taken into account towards data analysis of this endpoint. Only patients with measurements performed at the 3-month follow-up will be included in this analysis set. Specifically, the percentage of patients with an appropriate RV sensing at the 3-month follow-up will be determined.

All analyses are performed for patients with non-missing RV sensing data at the 3-month follow-up.

#### 24.2. Variables

CIP chapter 8.3.2.2.1 Rate of appropriate right ventricular sensing at 3-month follow-up

The parameter of interest  $Plexa_{Sensinq}$  is the rate of patients with appropriate sensing which will be calculated by  $Plexa_{Sensinq} = (Number of patients with appropriate sensing (Sensing_{app}))$  divided by number of patients with sensing measurements performed) \* 100%.

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | No | fu3_perf_rv_sens | Adequate RV sensing | nominal | Yes / No |

# 24.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

# 24.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 24.5. Descriptive Analyses

See general definitions in chapter 5.1.

#### 24.6. Hypotheses & Statistical Tests

Null hypothesis:  $H_{0\_Sensing}$ :  $Plexa_{Sensing} \le 93\%$ Alternative hypothesis:  $H_{A\_Sensing}$ :  $Plexa_{Sensing} > 93\%$ 

No multiplicity adjustment is performed for the secondary hypotheses. Thus a one-sided exact binomial test is carried out for the significance level 2.5%. Additionally, a two-sided 95% confidence interval for an exact binomial test is calculated.

<sup>&</sup>lt;sup>101</sup> analysis set Plexa SAR = Yes





# 25. Secondary EP: Rate appropriate RV pacing Plexa

# 25.1. Analysis set

All analyses are performed for the Plexa analysis set<sup>102</sup>.

CIP chapter 11.1 Statistical design, methods and analytical procedures

All endpoints are analysed per-protocol (PP), whereby the analysis sets are defined for each hypothesis separately.

<u>CIP chapter 8.3.2.2.2 Rate of appropriate right ventricular pacing at 3-month follow-up</u> Only the evaluation of the 3-month follow-up is taken into account towards data analysis of this endpoint. Only patients with measurements performed at the 3-month follow-up will be included in the endpoint.

All analyses are performed for patients with non-missing RV pacing data at the 3-month follow-up.

#### 25.2. Variables

CIP chapter 8.3.2.2.2 Rate of appropriate right ventricular pacing at 3-month follow-up
The parameter of interest  $Plexa_{Pacinq}$  is the rate of patients with appropriate pacing which will
be calculated by  $Plexa_{Pacinq} = (Number of patients with appropriate pacing (Pacing_{app}) divided
by number of patients with pacing measurements performed) * 100%. According to the
definitions provided in section 8.5.11, the pacing performance can be "adequate" or
"inadequate". If reason for inadequate performance is "No capture", the evaluation will not be
considered an endpoint-related event in case the underlying reason is a medical event (e.g.
hyperkalaemia, myocardial infarction or drug therapy).$ 

| Data file, identifier patient_display_id_full | Descri<br>ptive | Variable<br>name | Variable label, NEW prefix added to all labels "3mFU data: " | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| fu_3_month_<br>device_data | Yes | fu3_perf_rv_pac | Adequate RV pacing | nominal | Yes / No |

# 25.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 25.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

# 25.5. Descriptive Analyses

See general definitions in chapter 5.1.

#### 25.6. Hypotheses & Statistical Tests

Null hypothesis:  $H_{0\_Pacing}$ :  $Plexa_{Pacing} \le 93\%$ Alternative hypothesis:  $H_{A\_Pacing}$ :  $Plexa_{Pacing} > 93\%$ 

No multiplicity adjustment is performed for the secondary hypotheses. Thus a one-sided exact binomial test is carried out for the significance level 2.5%. Additionally, a two-sided 95% confidence interval for an exact binomial test is calculated.

<sup>&</sup>lt;sup>102</sup> analysis set Plexa SAR = Yes





# **Abbreviations**

ADE Adverse Device Effect

AE Adverse Event AF Atrial Fibrillation

CDMS Clinical Data Management System

CI Confidence Interval

CIP Clinical Investigation Plan
CIR Clinical Investigation Report

CRF Case Report Form

FU Follow-up

SADE Serious Adverse Device Event

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAR Statistical Analysis Report
SOP Standard Operating Procedure

SD Standard Deviation

